

| Official Title: | Geniculate Artery Embolization for Treatment of Knee Osteoarthritis |
|---|---|
| NCT Number: | NCT04379700 |
| Study Number: | 19-00370 |
| Document Type: | Study Protocol and Statistical Analysis Plan |
| Date of the<br>Document: | • May 6, 2025 |



#### Geniculate Artery Embolization for Treatment of Knee Osteoarthritis

| Principal Investigator: | Bedros Taslakian, M.D. |
|---|---|
| | Clinical Assistant Professor, Vascular and Interventional Radiology |
| | Director, VIR Research Program |
| | Department of Radiology, NYU Langone Health |
| | 550 First Avenue, 2 <sup>nd</sup> Floor, New York, NY, 10015 |
| | Email: Bedros.Taslakian@nyumc.org |
| | Phone: 929-434-1278 |
| Additional Investigators: | |
| | Jonathan Samuels, M.D. |
| | Associate Professor, |
| | Department of Internal Medicine, NYU Langone Health |
| | 333 East 38th Street, 4th Floor |
| | New York, NY 10016 |
| | Email: <u>Jonathan.Samuels@nyumc.org</u> |
| | Phone: 646-501-7400 |
| | - · - · |
| | Erin F. Alaia, M.D. |
| | Assistant Professor |
| | Department of Radiology, NYU Langone Health |
| | 560 1st Avenue, 2nd Floor |
| | Email: <u>Erin.Fitzgerald@nyulangone.org</u> Phone: 212-263-5941 |
| NYULMC Study Number: | s19-00370 |
| Funding Sponsor: | Department of Radiology |
| IND/IDE Number: | G190316 |
| Regulatory Sponsor: | Bedros Taslakian, M.D. |
| | Department of Radiology, NYU Langone Health |
| | Director, VIR Research Program |
| | 560 First Avenue, 2 <sup>nd</sup> Floor, New York, NY, 10015 |
| | Email: Bedros.Taslakian@nyumc.org; Phone: 212-263-5898 |
| Study Product: | Embozene™ Color-Advanced Microspheres |
| Study Product Provider: | Varian Medical Systems, Inc |
| ClinicalTrials.gov | NCT04379700 |
| Number | NO 1043/3/00 |

Initial version:04/16/2020Amended:19 Apr 2021Amended:31 January 2022Amended:07/06/2022Amended:02/08/2023Amended:06.25.2024Amended03.16.2025

Study number: s19-00370 Page ii

Version: 06.25.2024

#### **Statement of Compliance**

This study will be conducted in accordance with the Code of Federal Regulations on the Protection of Human Subjects (45 CFR Part 46), 21 CFR Parts 50, 56, 312, and 812 as applicable, any other applicable US government research regulations, and institutional research policies and procedures. The International Conference on Harmonisation ("ICH") Guideline for Good Clinical Practice ("GCP") (sometimes referred to as "ICH-GCP" or "E6") will be applied only to the extent that it is compatible with FDA and DHHS regulations. The Principal Investigator will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants. All personnel involved in the conduct of this study have completed Human Subjects Protection Training.

#### **Table of Contents**

| S | FATEMENT OF COMPLIANCE | II |
|---|---|---|
| LI | ST OF ABBREVIATIONS | VI |
| ΡI | ROTOCOL SUMMARY | 8 |
| S | CHEMATIC OF STUDY DESIGN | 10 |
| | KEY ROLES | |
| 1 | | |
| 2 | INTRODUCTION, BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE | 15 |
| | 2.1 BACKGROUND INFORMATION AND RELEVANT LITERATURE | |
| | 2.2 NAME AND DESCRIPTION OF THE INVESTIGATIONAL AGENT | |
| | 2.2.1 Preclinical Data | |
| | 2.2.2 Clinical Data to Date | |
| | 2.3 RATIONALE | |
| | 2.4 POTENTIAL RISKS & BENEFITS | |
| | 2.4.1 Known Potential Risks | |
| 3 | OBJECTIVES AND PURPOSE | 21 |
| | 3.1 PRIMARY OBJECTIVE | 21 |
| | 3.2 SECONDARY OBJECTIVES (IF APPLICABLE) | 22 |
| 4 | STUDY DESIGN AND ENDPOINTS | 22 |
| | 4.1 DESCRIPTION OF STUDY DESIGN | 22 |
| | 4.2 STUDY ENDPOINTS | |
| | 4.2.1 Primary Study Endpoints | |
| | 4.2.2 Secondary Study Endpoints Analysis | |
| 5 | STUDY ENROLLMENT AND WITHDRAWAL | 24 |
| | 5.1 INCLUSION CRITERIA | 24 |
| | 5.2 EXCLUSION CRITERIA | |
| | 5.3 VULNERABLE SUBJECTS | |
| | 5.4 STRATEGIES FOR RECRUITMENT AND RETENTION | |
| | 5.4.1 Use of DataCore/Epic Information for Recruitment Purposes | |
| | 5.5 DURATION OF STUDY PARTICIPATION | |
| | 5.6 TOTAL NUMBER OF PARTICIPANTS AND SITES | |
| | 5.7.1 Reasons for Withdrawal or Termination | |
| | 5.7.2 Handling of Participant Withdrawals or Termination | |
| | 5.8 PREMATURE TERMINATION OR SUSPENSION OF STUDY | |
| 6 | STUDY AGENT (STUDY DEVICE) AND/OR PROCEDURAL INTERVENTION | |
| | 6.1 STUDY DEVICE DESCRIPTION | |
| | 6.1.1 Acquisition | |
| | 6.1.2 Formulation, Appearance, Packaging, and Labeling | |
| | 6.1.3 Product Storage and Stability | |
| | 6.1.4 Preparation | |
| | 6.1.5 Dosing and Administration | |
| | 6.1.6 Route of Administration | |
| | 6.1.7 Duration of Therapy | |
| | 6.1.8 Device Specific Considerations | |
| | 6.2 STUDY PROCEDURAL INTERVENTION(s) DESCRIPTION | |
| | 6.2.1 Administration of Procedural Intervention Error! Bookmark not | аетіпеd. |

| Ve | sion: 06.25.2024 6.2.2 Procedures for Training of Clinicians on Procedural Intervention | 29 |
|---|---|---|
| 7 | STUDY PROCEDURES AND SCHEDULE | 30 |
| | 7.1 STUDY PROCEDURES/EVALUATIONS | 30 |
| | 7.1.1 Study Specific Procedures | |
| | 7.1.2 Standard of Care Study Procedures | |
| | 7.2 LABORATORY PROCEDURES/EVALUATIONS | |
| | 7.2.1 Laboratory Evaluations | |
| | 7.3 STUDY SCHEDULE | |
| | 7.3.1 Screening | |
| | 7.3.2 Enrollment/Baseline (Visit 2, Day -29 to -1)- In interventional radiology clinic | |
| | 7.3.3 Interventional visit (visit 3, Day 0) | |
| | 7.3.4 Follow-up Visits | |
| | 7.3.5 Withdrawal/Early Termination Visit | 34 |
| | 7.3.6 Unscheduled Visit | 34 |
| | 7.4 CONCOMITANT MEDICATIONS, TREATMENTS, AND PROCEDURES | 35 |
| | 7.5 RESCUE MEDICATIONS, TREATMENTS, AND PROCEDURES | 35 |
| | 7.6 PARTICIPANT ACCESS TO STUDY AGENT AT STUDY CLOSURE | 35 |
| 0 | ACCECCMENT OF CAFETY | 25 |
| 8 | ASSESSMENT OF SAFETY | 35 |
| | 3.1 SPECIFICATION OF SAFETY PARAMETERS | 35 |
| | 8.1.1 Definition of Adverse Events (AE) | 36 |
| | 8.1.2 Definition of Serious Adverse Events (SAE) | |
| | 8.1.3 Definition of Unanticipated Problems (UP) | 36 |
| | 3.2 CLASSIFICATION OF AN ADVERSE EVENT | |
| | 8.2.1 Severity of Event | 37 |
| | 8.2.2 Relationship to Study Device | 37 |
| | 8.2.3 Expectedness | 38 |
| | 3.3 TIME PERIOD AND FREQUENCY FOR EVENT ASSESSMENT AND FOLLOW-UP | |
| | 3.4 REPORTING PROCEDURES – NOTIFYING THE IRB | 39 |
| | 8.4.1 Adverse Event Reporting | 39 |
| | 8.4.2 Serious Adverse Event Reporting | 39 |
| | 8.4.3 Unanticipated Problem Reporting | 39 |
| | 8.4.4 Reporting of Pregnancy | 40 |
| | 3.5 REPORTING PROCEDURES - NOTIFYING THE STUDY SPONSOR | |
| | 3.6 REPORTING PROCEDURES – NOTIFYING THE FDA | 40 |
| | 3.7 STUDY HALTING RULES ERROR! BOOKMARK NOT DE | FINED. |
| | 3.8 SAFETY OVERSIGHT | 41 |
| 9 | CLINICAL MONITORING | 42 |
| 10 | STATISTICAL CONSIDERATIONS | 42 |
| | 10.1 STATISTICAL AND ANALYTICAL PLANS (SAP) | 42 |
| | 10.2 STATISTICAL HYPOTHESES | 42 |
| | 10.3 ANALYSIS DATASETS | |
| | 10.4 DESCRIPTION OF STATISTICAL METHODS | |
| | 10.4.1 General Approach | |
| | 10.4.2 Analysis of the Primary Endpoint(s) | |
| | 10.4.3 Analysis of the Secondary Endpoint(s) | |
| | 10.4.4 Safety Analyses | |
| | 10.5 SAMPLE SIZE | |
| 11 | SOURCE DOCUMENTS AND ACCESS TO SOURCE DATA/DOCUMENTS | |
| 12 | QUALITY ASSURANCE AND QUALITY CONTROL | 44 |
| 13 | ETHICS/PROTECTION OF HUMAN SUBJECTS | 45 |
| | 13.1 ETHICAL STANDARD | 45 |

| Study num | lber: s19-00370 | Page v |
|---|---|---|
| Version: 0 | * | |
| 13.2 | Institutional Review Board | |
| 13.3 | | |
| 13.3 | | |
| 13.3 | | |
| | PARTICIPANT AND DATA CONFIDENTIALITY | |
| | Research Use of Stored Human Samples, Specimens, or Data | |
| 13.5 | FUTURE USE OF STORED SPECIMENS | 46 |
| 14 DA | TA HANDLING AND RECORD KEEPING | 47 |
| 14.1 | DATA COLLECTION AND MANAGEMENT RESPONSIBILITIES | 47 |
| 14.2 | STUDY RECORDS RETENTION | 47 |
| 14.3 | PROTOCOL DEVIATIONS | |
| 14.4 | PUBLICATION AND DATA SHARING POLICY | 48 |
| 15 STL | IDY FINANCES | 48 |
| 15.1 | FUNDING SOURCE | 48 |
| 15.2 | COSTS TO THE PARTICIPANT | 48 |
| 15.3 | PARTICIPANT REIMBURSEMENTS OR PAYMENTS | 49 |
| 16 STL | IDY ADMINISTRATION | 49 |
| 16.1 | STUDY LEADERSHIP | 49 |
| 17 COI | NFLICT OF INTEREST POLICY | 49 |
| | ERENCES | |
| 19 ATT | ACHMENTS | 51 |
| | HEDULE OF EVENTS ERROR! BOOKMARK NOT | |

#### **List of Abbreviations**

| AE | Adverse Event/Adverse Experience |
|-------|-----------------------------------------------------|
| CFR | Code of Federal Regulations |
| CRF | Case Report Form |
| CSOC | Clinical Study Oversight Committee |
| CVA | Cerebrovascular accident |
| DCC | Data Coordinating Center |
| DHHS | Department of Health and Human Services |
| DSMB | Data and Safety Monitoring Board |
| DFU | Direction for Use |
| eCRF | Electronic case report form |
| FFR | Federal Financial Report |
| FWA | Federal wide Assurance |
| GCP | Good Clinical Practice |
| HIPAA | Health Insurance Portability and Accountability Act |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IRB | Institutional Review Board |
| ISM | Independent Safety Monitor |
| MOP | Manual of Procedures |
| MR | Magnetic Resonance |
| N | Number (typically refers to participants) |
| NIH | National Institutes of Health |
| OHRP | Office for Human Research Protections |
| OHSR | Office of Human Subjects Research |
| OA | Osteoarthritis |
| PI | Principal Investigator |
| PMMA | Polymethylmethacrylate |
| QA | Quality Assurance |
| QC | Quality Control |
| SAE | Serious Adverse Event/Serious Adverse Experience |
| SOP | Standard Operating Procedure |
| TP | Treating physician |

Study number: s19-00370 Version: 06.25.2024 Page vii

| US | United States |
|-------|----------------------------------------------------------------|
| UP | Unanticipated problem |
| VAS | Visual analog scale |
| WOMAC | Western Ontario and McMaster Universities Osteoarthritis index |
| WOMRS | Whole-Organ Magnetic Resonance Imaging Score |


### **Protocol Summary**

| Title | Genicular Artery Embolization for Treatment of Knee Osteoarthritis (OA) |
|---|---|
| Short Title | Geniculate Artery Embolization for Treatment of Knee Osteoarthritis |
| Brief Summary | Single-arm, single-center, no sham or placebo, prospective pilot trial designed to evaluate the feasibility and safety of transcatheter arterial embolization in patients with knee OA. Eligible participants will receive geniculate artery embolization using Embozene <sup>TM</sup> Color-Advanced Microspheres. Patients will be followed up for a total of 12 months. |
| Objectives | Primary objective: to determine the effectiveness of genicular artery embolization in reducing knee pain at 3-months post intervention in patients with knee OA. This will be assessed by evaluating the clinical success rate defined as at least 50% reduction in Western Ontario and McMaster Universities Osteoarthritis index (WOMAC) pain score from pre-intervention baseline to follow-up visit at 3 months post-intervention without an increase in baseline incidence of pain medication use or intra-articular injection. The WOMAC Score will be calculated from the Knee injury and Osteoarthritis Outcome Score (KOOS) score. Secondary objectives: To evaluate the safety of genicular artery embolization To determine whether transcatheter arterial embolization improves OA-related knee symptoms and quality of life. |
| Methodology | Prospective, single-arm, single-center, no sham or placebo, pilot study |
| Endpoint | Primary endpoint: WOMAC pain score at 3-months post intervention. Secondary endpoints: - Rate, type, causality, and severity of adverse events - WOMAC pain score at 1-,12-, and > 12-months post intervention - Pain visual analog scale (VAS) - WOMAC knee stiffness and physical function scores at 1, 3, 12 months |
| Study Duration | 3 years |
| Participant Duration | Each individual subject will be enrolled for approximately 13 months to complete all study visits from the initial screening visit to last follow up at 12-months post intervention. Participants that completed the 12 months visit by August 31, 2024 will be invited to participate in longer follow up (18 months – 48 months follow-up). |
| Population | 40 patients, age 30-80, any gender, with grade 2,3, or 4 (in select subjects with no bone deformity) knee OA on the most recent knee radiographs obtained within 6 months of intervention |

Study number: s19-00370 Version: 06.25.2024

| Study Sites | Single center: NYU Langone Health Hospitals |
|---|---|
| Number of participants | Data from 40 patients will be required The study would accrue 50 patients to account for an attrition rate of 20% |
| Description of Study<br>Agent/Procedure | Embozene™ Color-Advanced Microspheres are spherical, tightly calibrated, biocompatible, non-resorbable, hydrogel microspheres coated with an inorganic perfluorinated polymer used for embolization. |
| Key Procedures | Transcatheter arterial embolization of one or more genicular artery(ies) using<br>Embozene™ Color-Advanced Microspheres |
| Statistical Analysis | The primary objective is to assess the clinical success rate, which will be summarized in terms of the observed proportion of patients manifesting a positive response and a two-sided exact 95% confidence interval (CI) per the Blyth-Still-Casella method (reference). The treatment will be declared a success if the data support the conclusion that at least 75% of treated patients show a positive response. |

### Schematic of Study Design



### Schedule of Activities

| Visit # | Visit 1* | Visit2* | Visit 3 | Visit 4** | Visit 5# | Visit 6# | Visit 7# | Visit 8*** |
|---|---|---|---|---|---|---|---|---|
| Visit Description | Screening | Baseline | Intervention | 1-day<br>follow-up | 1-month<br>follow-up | 3-month<br>follow-up | 12-month<br>follow-up | >12<br>months |
| Eligibility screen | × | | | | | | | |
| Informed consent | × | | | | | | | |
| Demographics | | × | | | | | | |
| Medical history | | × | | | | | | |
| Adverse Events | | | | × | × | × | × | × |
| Physical exam | | × | | × | × | × | × | × |
| Medication History | | × | | | × | × | × | × |
| Pain VAS** | | × | | | × | × | × | × |
| KOOS score | | × | | | × | × | × | × |
| EQ-5D-5L scale | | × | | | × | × | × | × |
| Previous treatments | | × | | | × | × | × | × |
| Venous blood draws | | # <b>X</b> | # <b>X</b> | | × | × | × | × |
| Urine samples | | × | | | × | × | × | × |
| Knee MRI | | × | | | | ׳ | | |
| Knee radiograph | | $X^2$ | | | | | | |
| Genicular artery | | | × | | | | | |
| embolization | | | | | | | | |
| <ol> <li>If not previously available (i.e.,</li> </ol> | y available (i.e. | | recent knee MRI within 3 months of screening); if MRI cannot be obtained on the | onths of scre | ening); if MRI | cannot be obta | ained on the | 4 |

- If not previously available (i.e., recent knee MKI within 3 months of screening); if MKI cannot be obtained on the same day due to subject preference and/or MRI scheduling related reasons, MRI can be performed anytime between the baseline visit and intervention visit <u>.</u>
  - If not previously available (i.e., recent knee radiograph within 6 months of screening). Can be performed on a separate day based on appointment availability or subject's preference. 4
    - Post-procedural MRI can be done on a separate day of visit 6 based on appointment availability and subject's preference as long as it's performed within the timeframe of 3month +/- 10 days. က်
- \* Visit 1 and 2 can be combined based on subject preference. In that case, procedures listed in visit 2 will be performed after signing informed consent on the same day.
- \*\* Visit 4 (1-day follow-up) dates range can be +3 days (phone call, telemedicine, or in-person IR clinic visit determined by
- subject's preference and need for physical examination)
  \*\*\* Visit 8. Optional visit for participants who completed 12 month follow up by August 31, 2024 (by invitation, voluntary, and after obtaining informed consent for this visit). This visit can be performed at any time interval within 18 months – 48 months


Version: 06.25.2024

post procedure. This visit can be performed by sending the questionnaire by a safe email and participants can email it back to research coordinator or PI OR by a phone call performed by research coordinator,


# 1, 3, 12-month follow-up dates range can be +/- 10 days

## The pre-procedural blood work can be done on the day of the procedure prior to performing the procedure based on subject's preference.

Version: 06.25.2024

### **Key Roles**

Principal Investigator (PI): Will be one of two interventional radiologists performing the procedure. Will be responsible for study integrity, data monitoring, data collection, statistical analysis, and manuscript writing.

### Bedros Taslakian, MD

Clinical Assistant Professor of Radiology

Director, Vascular and Interventional Radiology Research Program

Department of Radiology, NYU Langone Heath

550 First Avenue, 2nd Floor, New York, NY 10015

Phone: 929-434-1278

Email: Bedros.Taslakian@nyumc.org

Co-PI: Co-investigator involved in recruiting patients and conducting the clinical assessment for knee osteoarthritis

Jonathan Samuels, M.D

Associate Professor

Department of Internal Medicine, NYU Langone Orthopedic Center

333 East 38th Street, 4th Floor

New York, NY 10016

Email: Jonathan.Samuels@nyumc.org

Co-PI: Co-investigator (musculoskeletal radiologist) conducting the imaging assessment

### Erin F. Alaia, MD

Assistant Professor

Department of Radiology, NYU Langone Health

560 1st Avenue, 2nd Floor

Email: Erin.Fitzgerald@nyulangone.org

Phone: 212-263-5941

### Research Coordinator:

Biostatistician: Will be responsible for conduction statistical analysis

James Babb, PhD

Department of Radiology, NYU Langone Health

660 First Avenue

New York, NY 10016

Phone: 212-263-3782

Email: James.Babb@nyulangone.org


Introduction, Background Information and Scientific Rationale

## 2.1 Background Information and Relevant Literature

Knee OA is common and major cause of pain and disability. Its prevalence is rising due to an aging population and the high prevalence of obesity 1]. Radiographically confirmed symptomatic knee OA affects approximately 3.8% of people worldwide, and knee and hip OA ranked as the 11th highest contributor to global disability [2]. Disabling symptoms of knee osteoarthritis are seen in an approximately 10 % of people over 55 years old [3]. Therefore, the prevalence and burden of knee OA presents a major challenge for health systems globally [2].

joint injury, bone and joint shape, muscle strength and mass, obesity, gender, metabolic factors, nutrition and vitamin factors, bone density, Knee OA is a complex, multifactorial disease with no known cure. Risk factors for knee OA include psychological health and occupation [4, 5]. Treatment seeks

to manage symptoms, but adequate symptom control can be difficult to achieve [4-6]. Evidence-based treatment options for knee OA include intralimitations [8, 9]. On the other hand, moderate knee OA resistant to nonsurgical options, yet not severe enough to warrant joint replacement, does not have an optimal therapy. Therefore, there is still a need to develop an effective, minimally invasive and safe treatment for moderate OA of the inflammatories for minor symptoms [7]. Total knee arthroplasty is generally reserved for those with severe joint disease, pain and functional articular corticosteroids, exercise, education, weight management, and oral medications such as acetaminophen and non-steroidal anti-

structural damage, inflammation and pain [10]. Angiogenesis is blood vessel overgrowth from pre-existing vasculature and is essential for growth, development and tissue repair [10]. However, in OA, angiogenesis increases in articular cartilage, synovium, meniscus, and osteophytes, and at symptoms of OA [10]. Angiogenesis inhibitor treatment decreased pain-related behavior in animal models [11]. The mechanism of symptomatic aneural structures such as articular cartilage and meniscus is thought to contribute to OA pain through chemical and mechanical stimulation of the osteochondral junction [11-15]. Because angiogenesis is accompanied by sensory nerve growth, perivascular nerve growth into normally An in-depth understanding of OA pathophysiology is still emerging [1]. Recently, angiogenesis has been implicated in OA by contributing to newly formed nerves. Modifying angiogenesis and associated nerve growth is a potential treatment pathway to affect the pathogenesis and relief is unclear but could include reduced synovitis, reduced periarticular innervation and nociception, and maintaining the integrity of the osteochondral junction [10, 11].

grade 2 in 18% of the patients, grade 3 in 43%, and grade 4 in 40%. Technical success was achieved in 100% of the subjects. The WOMAC total A recent study by Padia S et al evaluated the safety and effectiveness of GAE in patients with knee OS (grades 2, 3, 4). Knee OA severity was and VAS pain scores decreased by 61% and 67% at 12 months from a median baseline of 52 (of 96) and 8 (of 10), respectively. Twenty-seven patients (68%) had a reduction of ≥50% in both WOMAC total and VAS pain scores [32].

The WOMAC questionnaire is a widely used, disease-specific measure for knee OA. It includes 24 questions on daily activities: five regarding stiffness, 0-8; and physical function, 0-68. For each question in each of the three categories (pain, stiffness, and physical function) patients receive the following points: 0 for no symptoms, 1 for mild, 2 for moderate, 3 for severe, and 4 for extreme symptoms. Higher scores on the pain, two regarding stiffness, and 17 regarding physical function; possible score ranges for each subset of items are as follows: pain, 0-20; WOMAC indicate worse pain, stiffness, and functional limitation [16]. The Whole-Organ Magnetic Resonance Imaging Score (WORMS) in patients with knee OA provides multi-feature, whole-organ assessment of the knee in OA using conventional magnetic resonance imaging (MRI), and shows high inter-observer agreement among trained readers [17]. Wholeorgan assessment could help discriminate different patterns of intra-articular involvement in OA; detect early, potentially preclinical, stages of OA;


functional integrity of the knee and/or potentially involved in the pathophysiology of OA. It scores each of these features with a sufficient number of treatment response in patients with established OA. It takes into account a variety of features that are currently believed to be relevant to the identify structural risk factors for developing clinical OA; or increase scope and sensitivity to change for monitoring disease progression and increments to allow detection of what are speculated to be clinically relevant changes.

## 2.2 Name and Description of the Investigational Agent

The investigation agent (device) in this trial is Embozene™ Color-Advanced Microspheres.

target tissue. They are available in prefilled syringes in a range of sizes suitable for embolic therapy. The microspheres are compressible to enable Embozene™ Color-Advanced Microspheres are spherical, tightly calibrated, biocompatible, nonresorbable, hydrogel microspheres coated with an smooth delivery through the indicated delivery catheter and color-coded by size to allow for easy identification. In this trial, we intend to use 250 inorganic perfluorinated polymer (Polyzene™-F). The microspheres intended to occlude vasculature for the purpose of blocking blood flow to a um microspheres (range of microsphere sizes is 250 µm ± 50 µm as per manufacturer, prefilled in yellow syringes).

approximately 7 ml. Prefilled syringes of Embozene™ Color-Advanced Microspheres are packaged in a sterile, sealed tray with a peel-away lid. Embozene™ Color-Advanced Microspheres are supplied in a 20 ml syringe prefilled with 2 ml of product suspended in a non-pyrogenic, sterile transport solution of physiological saline. The total volume of Embozene™ Color-Advanced Microspheres including transport solution is The label indicates the specific size of the microspheres contained in the syringe.

Embozene™ Color-Advanced Microspheres are intended for embolization of arteriovenous malformations and hypervascular tumors, including uterine fibroids and hepatoma, and for embolization of prostatic

indications (FDA approved for treatment of benign prostatic hyperplasia; FDA 510(K) # K180102; 510(k) premarket notification of intent to market arteries for symptomatic benign prostatic hyperplasia. This device is not intended for neurovascular use. The device is FDA approved for above the device FDA 510(k) # K141209)

There are no known chemical interactions between Embozene™ Color-Advanced Microspheres and pharmaceuticals.

Additionally, for labeling with Magnetic Resonance (MR) compatibility, the proposed Embozene TM Color-Advanced Microspheres were assessed and met requirements in the Guidance for Industry and Food and Drug Administration Staff Establishing Safety and Compatibility of Passive Implants in the MR Environment. Embozene TM Color-Advanced Microspheres are labeled MR safe in the device Direction for Use (DFU) attachment 1]

IDE for the purpose of this study was obtained from the FDA (IDE approval # G190316. Approval letter provided [attachment 2].

FDA documents of the device under investigation for approved indications and device DFU are attached to this IRB protocol [attachments 3,4].

FDA reviewed the supplement of IDE application to expand study for significant risk device proposing the addition of 21 patients. FDA has determined sufficient data to support expansion of human clinical trial; this means there are no subject protection concerns that preclude expansion of the investigation. Approved to expand study. Limit 1 US institution and 50 US subjects. [attachment G190316-S003. Letter.EPEX.APPR]


2.2.1 Preclinical Data

that using the device for geniculate artery embolization (for treatment of knee OA) does not require additional bench, biocompatibility, sterilization, requirements for its intended use. As the device received FDA approval for additional indications lately (prostate artery embolization), we believe or pre-clinical animal testing beyond what was required for the reference device. All existing testing provided in the Non-clinical tests performed on the Embozene Microspheres, reference device, provide reasonable assurance that the proposed device has been designed and tested to assure conformance to the previous Embozene Microspheres premarket submissions remains applicable. Biocompatibility testing provided in the previous Embozene Microspheres premarket notification included: cytotoxicity, sensitization, irritation, subchromosome aberration, in-vivo micronucleous assay), implantation, hemocompatibility (hemolysis, partial thromboplastin time, platelet/leukocyte acute and sub-chronic systemic toxicity, systemic toxicity- material mediated pyrogenicity, genotoxicity (bacterial mutagenicity, in-vitro counts). All tests passed, indicating that the device materials are biocompatible for its intended use.

inspection, Ph of transport solution, osmolality of transport solution, microsphere suspension, catheter compatibility, and elution test. all tests Performance testing provided in the previous Embozene Microspheres premarket notification included: microsphere size distribution, visual passed demonstrating the device meets the predetermined performance requirements. Published literature on preclinical animal studies assessed the biocompatibility, safety, and efficacy of Embozene Microspheres in comparison with inflammatory reactions. The results demonstrate a similar biological tissue response between the Embozene Microspheres and the Embosphere distribution characteristics, inflammation and recanalization, impact on inflammatory tissue and foreign body reaction, and immunohistochemical the Embosphere predicate and other embolization devices. The devices were evaluated in a porcine kidney model to determine arterial predicate device which supports substantial equivalence [18].

A study by Stampfl et al, evaluated the inflammatory response and recanalization after embolization with the embolic agent based on a core and shell design with a hydrogel core of polymethylmethacrylate (PMMA) and a Polyzene-F nanoscale coating in a porcine kidney model [19]. It demonstrated good biocompatibility of the embolic material. As in other spherical embolic agents, recanalization can occur to some degree. Additionally, for labeling with MR compatibility, the proposed Embozene Microspheres were assessed and met requirements in the Guidance for Industry and Food and Drug Administration Staff Establishing Safety and Compatibility of Passive Implants in the MR Environment.

### 2.2.2 Clinical Data to Date

Embozene Microspheres have been already investigated in several clinical studies. Stampfl U et al, investigated the safety and efficacy of uterine Polyzene F-coated hydrogel microspheres for uterine artery embolization resulted in good dominant and overall tumor infarction in most patients, reduction rates and significant improvements of clinical symptoms and quality-of-life scores during follow-up [20]. Sneets el al, demonstrated that embolization with Embozene microspheres is a safe procedure. Its efficacy is demonstrated by high fibroid devascularization and volume artery embolization using narrow-size-range polyphosphazene-coated hydrogel microspheres. Results demonstrated that uterine artery with corresponding improvement of symptoms [21].


Page 18 Study number: s19-00370 Embolization of the geniculate artery was also investigated for the treatment of recurrent hemorrhage after hip and knee arthroplasty. Kalmar et al demonstrated 100% technical success rate, no procedure-related complications, and effectiveness in patients without underlying coagulopathy in preventing recurrences of spontaneous recurrent hematoma or hemarthrosis of the hip and the knee [22]

abnormal branches of the genicular artery using imipenem and cilastatin sodium or 75 µm Embozene microsphere. WOMAC pain and function scores improved substantially at 1, 4, and 12 months post procedure. No major adverse events occurred. One participant had a moderate Recently, embolization of the geniculate artery was evaluated for the treatment of knee OA. Okuno et al, investigated the effects of embolizing abnormal blood vessels in people with mild to moderate knee OA [6]. Fourteen participants received transcatheter arterial embolization of subcutaneous hemorrhage at the puncture site that resolved within 1 week. In a follow-up study, Okuno et al, described the safety and efficacy of transcatheter arterial embolization in 72 patients with mild to moderate radiographic knee OA [23]. Clinical outcomes were evaluated at 1, 4, and 6 months and then every 6 months for a maximum of 4 years. Mean WOMAC pain scores significantly decreased from baseline to 1, 4, 6, 12, and 24 months after treatment (12.1 vs 6.2, 4.4, 3.7, 3.0, and 2.6; all P < .001). The WORMS score was evaluated at baseline and at 2 years after embolization in 35 knees and showed significant improvement of synovitis vs baseline (P < .0016) and no osteonecrosis or other evidence indicating aggressive progression of degenerative changes. There were no major adverse events related to the procedures. Specifically, there was no incidence of tissue necrosis, dermal ulcers, or peripheral paresthesia in any embolized territory during the follow-up period. Moderate subcutaneous hemorrhage at the puncture site in 12 patients resolved within 1 week. Four of seven patients treated with Embozene showed transient cutaneous color change on the treated knee, which resolved spontaneously within 1 A recent study by Bagla et.al, showed improvement in the pain scores in 20 patients with knee osteoarthritis. The mean VAS improved from 76 mm  $\pm$  14 at baseline to 29 mm  $\pm$  27 at 6-month follow-up (P <.01). The mean WOMAC score improved from 61  $\pm$  12 at baseline to 29  $\pm$  27 at 6-month follow-up (P < .01). Self-limiting skin discoloration occurred in 65% patients and 10% of patients developed transient plantar sensory paresthesia.

### 2.3 Rationale

The rational is based on a recent article by Okuno Y et al [23]. "The hallmark symptom of knee OA is pain. This is the symptom that drives individuals treatment, including nonpharmacologic, pharmacologic, and surgical approaches. Severe and end-stage knee OA is successfully treated with joint to seek medical attention and contributes to functional limitation and reduced quality of life [24, 25]. The alleviation of pain is the main motivation for replacement surgery, but effective management of mild to moderate radiographic knee OA refractory to conservative treatment can be difficult." 'Although OA was viewed as a "wear-and-tear" disease for many decades, it is now generally accepted to be a low-grade inflammatory disease of to its maintenance [11]. The new increased vascular network provides inflammatory cells access to the synovium and other joint tissues and promotes additional hyperplasia and inflammation in other vessels, leading to bone and cartilage destruction [27]. In addition, studies on OA have shown that synovial joints and a biomechanical whole-organ disease [26]. Angiogenesis is believed to contribute to the genesis of inflammation and particularly angiogenesis may contribute to chronic pain by enabling the growth of new unmyelinated sensory nerves along their path [12, 15]." The current study seeks to determine whether transcatheter arterial embolization of abnormal neovasculature arising from the genicular arterial branches is safe and effective in the treatment of mild-to-moderate knee OA.


Version: 06.25.2024

### Potential Risks & Benefits

### 2.4.1 Known Potential Risks

Potential adverse events related to the use of the device from the device from the device insert of directions for use (DFU) [attachment 1] and recent literature [6, 23]:

- Possible adverse events:
- Incomplete occlusion of vascular beds or territories may give rise to the possibility of post-procedural development of alternative vascular pathways, recanalization, or recurrence of symptoms
- Post-embolization syndrome including fever, malaise, headache, and myalgia (body aches)
- Transient, self-resolving cutaneous purpura / skin color change
- Transient plantar or peripheral sensory paresthesia
- Synovitis related symptoms including pain, stiffness or limited joint mobility
- Rare adverse events:
- Allergic reaction and foreign body reactions (e.g., pain, rash, fever, inflammation)
  - Capillary bed saturation and tissue damage
- Infection
- Neurological deficits
- Pulmonary embolization
- Thrombosis
- Undesirable reflux, passage/migration or placement of Embozene™ Microspheres, resulting in non-target embolization, ischemia, and / or ischemic infarction.
- Non-target embolization to lower extremity vasculature resulting in vascular thrombosis and limp threatening ischemia
- Vessel or lesion rupture
- Tissue necrosis
- Dermal ulcer
- Fendon or ligament rupture
- Osteonecrosis (rare- not reported in prior studies)
- Joint infection (rare- not reported in prior studies)
- Very rare adverse events:
- Cerebrovascular accident (CVA)

Potential adverse events associated with angiography and catheterization of vessels include:

- Nausea, vomiting, and/or allergic reaction anaphylaxis due to iodinated contrast used during embolization procedure (less possible)
  - Contrast-induced renal dysfunction (less possible)
- Access site-related adverse events: bleeding, infection, hematoma formation, arteriovenous fistula, pseudoaneurysm (rare)


Vessels catherization associated adverse events: injury to catheterized vessels including vessel perforation, dissection, vasospasm, or

- Vessels cattletization associated adverse events, injury to thrombosis (rare)
- Infection (rare)

Potential adverse events associated with radiation exposure due to use of knee radiograph and fluoroscopy

- Deterministic radiation risks: Radiation-induced injuries to the skin and underlying tissues, which occur shortly after the exposure (rare)
- Stochastic radiation risks: Radiation-induced malignancy which may occur later in life (rare)

Potential adverse events associated with MRI knee:

- Discomfort (possible)
- Anxiety or claustrophobia (less possible)
- Peripheral nerve stimulation casing tingling or twitching (rare)
- Injury and burns related to metals (very rare, particularly with the MR screening performed prior to entering MR zone and subjects with contraindications to MR will be excluded from the study)
- Pacemaker dysfunction (very rare; subjects with pacemakers will be excluded from the study)
- Skin burns (very rare)
- Tinnitus and hearing loss (very rare)
- Quench (very rare)

Potential adverse events associated with moderate sedation during procedure:

- Over sedation (less possible)
- Nausea, vomiting, and/or allergic reaction to medications / anaphylaxis (rare)
- Respiratory failure, myocardial infarction, and death (rare)

Potential risks associated with study enrollment and ancillary study procedures:

- Discomfort due to blood draws required for the study (possible)
- Minor local discomfort due to the pressure of the ultrasound transducer on the skin during arterial access (possible)
  - Inconvenience at having to return for follow-up visits (possible)
- Discomfort, Thrombophlebitis, bruising, bleeding, blood clot, presyncope or syncope (i.e. fainting) due to blood draws required for the study (less possible)
- Psychological discomfort from clinical trial enrollment and completing study questionnaires (less possible)
  - Infection from blood draw for lab tests (rare)
- Loss of confidentiality of medical records (rare)

### Risk minimization:

The GAE procedure will be performed by fellowship-trained interventional radiologists who have expertise in endovascular techniques, particularly in selective catheterization and transcatheter embolization techniques.


Analgesia during the procedures will be provided using conscious sedation if subject opted to receive conscious sedation. The risks of conscious sedation will be minimized by continuous monitoring of heart rate, blood pressure, oxygen saturation, and cardiac rhythm.

background radiation and significantly less than that of a cardiac catheterization (reference: Phys Med. 2009 Mar; 25(1):25-30). Radiation exposure will be minimized to subjects under the principal of 'as low as reasonably achievable' (ALARA). For example, fluoroscopy will be performed with The dose area product projected for the procedure is thought to be around 30-75 gray/cm2. The effective radiation dose is approximately 0.003 the lowest acceptable exposure for the shortest time necessary to perform the procedure (genicular artery embolization). Methods to reduce mSv from the x-ray of the knee if needed and a mean of 3.0 to 12 mSv from angiography of the lower extremity which is about 2-4 years of radiation-related adverse events include, but not limited to, tight collimation, use of pulsed fluoroscopy, and judicious image acquisition.

be minimized by administration of local anesthesia into the overlying skin and adjacent tissues. Catheter access into the appropriate artery may be Sterile instruments with a sterile technique will be used to minimize infection risk at the arterial access site. The arterial access site discomfort will performed using ultrasound-guided arterial puncture to prevent inadvertent vessel puncture with subsequent bleeding. Real-time fluoroscopic monitoring of all catheter/wire manipulations will be used to prevent vascular injury.

Cone beam CT, which provides cross sectional anatomic detail prior to embolization, will be available to the operating interventional radiologist. This angiographic technique can mitigate the risk of non-target embolization. The intent of this technique, as well as meticulous angiographic technique will be used to minimize the risk of non-targeted embolization, that could lead to skin or soft tissue/muscle injury. The subject will be monitored for the risk of an allergic response to iodinated contrast. To minimize the risk of renal dysfunction there will be use of non-ionic contrast agents, and appropriate pre-procedure hydration, when necessary. Subjects who report an allergic reaction to iodinated contrast will be pre-medicated as per routine allergy prophylaxis per standard of care.

### 2.4.2 Known Potential Benefits

There is no guarantee of benefit to any subject. Potential benefits to the subjects from participating in the study, based on prior clinical data available in the literature [6, 23] are:

- Knee pain reduction
- Physical function improvement
- Synovitis reduction

Other potential benefits under investigation:

- Quality of life improvement
- Delay in progression of disease (i.e. knee OA)

### 3 Objectives and Purpose

### 3.1 Primary Objective

The primary objective of the study is to determine the effectiveness of genicular artery embolization in reducing knee pain at 3-months post intervention in patients with knee OA. This will be assessed by evaluating the clinical success rate defined as at least 50% reduction in WOMAC


pain score from pre-intervention baseline to follow-up visit at 3 months post-intervention without an increase in baseline incidence of pain medication use or intra-articular injection.

### Secondary Objectives

The secondary objectives of the study are to determine whether genicular artery embolization is effective in improving

- Knee pain using an electronic VAS at 1-, 3-, and 12-months (and final 18-48 months visit) post intervention
  - Knee pain using WOMAN pain score at 1- and 12-months (and final 18-48 months visit) post intervention
- knee stiffness using the WOMAC knee stiffness score at 1-, 3-, and 12- months (and final 18-48 months visit) post intervention લં છં
- Physical function using the WOMAC function score at 1-, 3-, and 12- months (and final 18-48 months visit) post intervention
  - Self-reported quality of life using EQ-5D-5L scale at 1-, 3-, and 12- months (and final 18-48 months visit) post intervention [28] Synovitis on MRI at 3 months post intervention
  - 4. 7. 0.

Other secondary objectives are to assess

- Feasibility / technical success defined as successful selective catheterization of target vessel(s) and embolization from at least one feeding artery of the knee joint (with the embolization endpoint defined as suppression or reduction in the filling of (and therefore blood flow in) abnormal vessels visible on angiography.
- Reduction in frequency of pain medication usage over 30-day period assessed at baseline and at 1, 3, and 12 months follow-up visits post intervention (acetaminophen, over the counter NSAIDs, prescription NSAIDs, opioids) ď
- Reduction in frequency of knee injection therapy over 12-month period (assessed at baseline and at 12-month follow-up visit post intervention) რ
- Reduction in frequency of need for physical therapy over 12-month period (assessed at baseline and at 12-month follow-up visit post intervention) 4
- Safety evaluated by cumulative rates of adverse events (AE), as well as type and severity of each adverse event. 5.

## Study Design and Endpoints

## 4.1 Description of Study Design

This study is a single-center, single arm, no sham or placebo, open label, prospective pilot study designed to evaluate the safety and feasibility of geniculate arteries in the affected knee using 250 µm Embozene microspheres. If both knees are affected, the knee with the higher pain score on geniculate artery embolization for the treatment of knee OA. Enrolled patients will receive angiography and embolization of the one or more electronic VAS will be targeted. The primary objective is to evaluate the effectiveness of geniculate artery embolization in reducing knee pain at 3 months. The primary objective will be evaluated by the clinical success rate. Clinical success is defined as at least 50% reduction in WOMAC pain score at 3-month follow up visit. 40 patients will be required for this study. The study would accrue 50 patients to account for an attrition rate of 20%.

Change in WOMAC pain score and pain VAS will be used as a measure of efficacy (i.e., pain reduction).

WOMAC questionnaire is a widely used, disease-specific measure for knee OA. It includes 24 questions on daily activities. WOMAC pain score includes five questions regarding pain (pain during walking, stair climbing, nocturnal, rest, weight bearing); each question will be scored suing the


osteoarthritis. This means that the KOOS questionnaires will be administered to patients during visits and the WOMAC score will be calculated from following points: 0 for no pain, 1 for mild, 2 for moderate, 3 for severe, and 4 for extreme pain. possible score ranges for pain are 0-20. For this purpose, WOMAC Score will be calculated from the Knee injury and Osteoarthritis Outcome Score (KOOS) score which was developed as an extension of the WOMAC score with the purpose of evaluating short-term and long-term symptoms and function in subjects with knee injury and the KOOS scores later at the time of data analysis. The electronic VAS is a horizontal line with no markings on the scale except "No pain" on the left (score: 0 mm) and "worst possible pain" on the representing "worst possible pain". In our study, subjects will be asked to mark their pain level on a paper VAS on study questionnaire form and will right end of the scale (score: 100 mm). Subjects mark the VAS to indicate their current pain level, with 0 mm representing "No pain" and 100 mm give a score between 0 to 100, which will be documented on the appropriate eCRF. All study variables will be collected on paper form [forms # 1-7 attached to this protocol] and study questionnaire forms (source documents) at the time of each clinic visit and transferred to eCRFs (TrialMaster; on NYU Langone secure servers) by the study coordinator or an investigator. The source documents (paper forms) will be placed in secure locked folders with study documents (such as signed consent forms). The data dictionary of TrialMaster will be similar to the attached forms, [attachment 5].

### 4.2 Study Endpoints

### 4.2.1 Primary Study Endpoints

The primary endpoint is WOMAC pain score at 3 months post intervention.

## .2.2 Secondary Study Endpoints Analysis

### Secondary efficacy endpoints are:

- WOMAC pain score at 1- and 12- months (and final 18-48 months visit) post intervention
- Pain electronic VAS at 1-, 3-, and 12- months (and final 18-48 months visit) post intervention
- Knee stiffness WOMAC score at 1-,3-, and 12- months (and final 18-48 months visit) post intervention
- Physical function WOMAC score at 1-, 3-, and 12- months (and final 18-48 months visit) post intervention 4
- Total WOMAC score at 1-,3-, and 12- months post intervention
- Self-reported quality of life using EQ-5D-5L scale at 1-, 3-, and 12- months (and final 18-48 months visit) post intervention. 6
  - 7- MRI findings at 3- months post intervention
- Pain medication usage at 1-, 3-, and 12- months (and final 18-48 months visit) post intervention
- Injection therapy requirements (hyaluronic acid or steroid) at 12- months (and final 18-48 months visit) post intervention
  - Physical therapy requirements at 12- months (and final 18-48 months visit) post intervention
    - 11- Feasibility / technical success
- 12- Laboratory findings at 1-, 3-, and 6- months (and final 18-48 months visit) post intervention

### Secondary safety endpoints are:

13- Number/rate, severity, and description of complications, adverse events, or poor outcomes that are secondary to the procedure, which will be summarized using counts and simple statistics (i.e., mean number of patients with complications.)


## Study Enrollment and Withdrawal

### 5.1 Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all the following criteria:

- 30-80 years of age of any gender and; Kellgren-Lawrence Grade 2, 3, or 4 (in select subjects who have no bony deformity)# knee OA on most recent knee radiograph obtained within 6 months of screening visit and;
- Knee pain resistant to conservative treatment for at least 3 months\* (anti- inflammatory drugs, acetaminophen, physical therapy, muscle strengthening, or intra- articular injection of hyaluronic acid and/or steroids); and რ
  - Moderate to severe knee pain: pain VAS ≥40 mm with 0 representing 'no pain' and 100 'the worst pain imaginable. If both knees meet inclusion criteria, the one with a higher VAS score will be chosen for the study (i.e., target knee). 4.
- Willing, able, and mentally competent to provide informed consent and complete study questionnaires in English. The Study questionnaire is validated in English. 5

pain score with no added risks. The scientific rational for adding these subjects with KL grade 4 (severe knee OA with no bone deformity) is based # A recent study by Padia S et al included subjects with KL grade 4 and published results showed, similar to other studies, clinical reduction in on recent literature data (Citation: JB JS Open Access. 2021 Oct-Dec; 6(4): e21.00085.)

\*3 months was chosen because this time interval is thought adequate for knee pain to be considered refractory to conservative care.

### Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

- Active systemic or local knee infection or;
  - Active malignancy or;
- Life expectancy less than 12 months or; ω. <del>4</del>.
- Prior ipsilateral knee surgery (within 3 years of baseline visit), arthroscopic surgery (within 6 months of baseline), total or partial knee replacement regardless of timing or;
  - psilateral knee intra-articular injection in the last 3 months or;
  - Rheumatoid arthritis, spondyloarthropathies, crystal disease, gout, pseudogout, or lupus, . 6. 7. 8
    - Pregnant during the study period or;
- Renal dysfunction as defined by serum creatinine >1.6 dl/mg or eGFR <60 on blood tests obtained within 30 days of procedure or;
  - Body weight greater than 200 Kg or;
- Uncorrectable coagulopathy (platelet count < 50,000, international normalized ratio >1.5 within 30 days of procedure; or 6.
  - Known history of contrast allergy resulting in anaphylaxis or; 7. 5.
- Known significant arterial atherosclerosis that would limit selective angiography and/or lower extremity symptoms thought to be secondary to arterial vascular disease (eg claudication, ischemic rest pain)
  - Post-traumatic knee (if trauma occurred within 12 months of baseline or was associated with fractures)
- known avascular necrosis in the target knee
- Contraindications to MRI such as such as claustrophobia, metallic fragment/implants, pacemaker.


### 5.3 Vulnerable Subjects

The study does not intend to recruit vulnerable subjects. The study will not recruit any children, pregnant women, fetuses, neonates, or prisoners.

## 5.4 Strategies for Recruitment and Retention

assess the medical record of potential subjects for eligibility and provide eligible participants with written information (i.e. study brochure) regarding Participants will be recruited at the study investigator or sub-investigator clinical practices (visit 1). A study investigator or sub-investigator will the study during the initial study visit [attachment 6] and obtain informed consent.

the Kellgren-Lawrence scale by a board certified, fellowship-trained musculoskeletal radiologist (Co-PI) [29]. Recruitment is expected to occur over 3 years. To achieve primary objective, data from 40 patients will be required and the study would accrue 50 patients to account for an attrition rate RB-approved study coordinator or co-investigator will guide interested people through written informed consent. knee X-rays will be graded with

medicine, and interventional radiology clinics and will be also disseminated on social media (e.g. Facebook, Twitter, blogging) to advertise for the study after IRB approval. The study brochure will include contact information for interested subjects to contact study coordinator and/or PI. Only NYULH individuals who are listed on the NYU Langone Health IRB-approved protocol will approach patients for consent. A study brochure will be provided for potential subjects [attachment 6]. The study brochure will also be available in NYULH rheumatology, orthopedics, family

Once enrolled, IRB-approved study coordinator will notify and remind participants about the visits.

Participation in the study is voluntary; no financial incentives will be offered.

## 5.4.1 Use of DataCore/Epic Information for Recruitment Purposes

generate a list of potential subjects with a diagnosis of knee OA and who meet eligibility criteria from the electronic medical system of NYULH. This study will utilize EPIC to identify subjects. DataCore will request a report after obtaining IRB approval. The report will be requested to

The VIR / Radiology research coordinator, Bedros Taslakian (PI), Akhilesh Sista (co-PI), and Jonathan Samuels (co-PI) will have access to EPIC search results. The list will be filtered to identify patients who meet eligibility criteria listed in this protocol.

The PHIs that will be extracted from the EPIC search will be patient's name, MRN, contact information, and name and contact information of the treating physician (TP). The dataset will be deleted after discontinuation, termination, or completion of the study.

Queries regarding eligible subjects will run during the course of the study once a month until discontinuation, termination, or completion of the

Once potential subjects have been identified, the study team will notify the TP that they have patients eligible to participate as follow:

Treating physician will be notified that the study team will contact potential subjects directly, by phone, email, or the MyChart portal.


If TP agrees to permit study team to directly contact potential subjects on behalf of TP, a study coordinator or investigator will inform the potential subjects about the study using standard language [attachments 7&8] and study brochure [attachment 6]

language attached to this protocol [attachments 7 and 8]. When sending recruitment information by email, SendSafe Secure email will be used to Patients will be contacted by email, the MyChart portal, MyChart recruitment tools through DataCore, and/or direct phone call using standard contact patients. Once contact is made, the IRB-approved study brochure or language included in the approved study brochure (if contact made by phone) will be used to communicate the reason they are being contacted and subjects will be asked if they are interested in participating in this specific study. Should the potential subjects agree, the study team will provide the subjects with information regarding the next steps for participation.

the study brochure. If patient agrees to participate, he will be scheduled for a clinic visit with one of the investigators (visit 1) to further discuss the coordinator or the PI at Bedros Taslakian@nyulangone.org or at the office number 212-263-5898. The contact information is also be available on If a subject requests information regarding opting out of further recruitment for all research, subjects will be directed to contact the VIR research study, complete the screening elements, and obtain informed consent. If a subject requests information regarding opting out of further recruitment for all research, subjects will be directed to contact study coordinator or have subjects contact research-contact-optout@nyumc.org or 1-855-777-7858.

## 5.5 Duration of Study Participation

Each subject will be enrolled in the study for approximately 13 months from the initial screening visit (visit 1; Day -30) until the last follow-up visit at 12 months post intervention (visit 7; Day 360)

## 5.6 Total Number of Participants and Sites

Data from 40 participant will be required and the study would accrue 50 patients to account for an attrition rate of 20%.

The study will be conducted only at NYULH Hospitals. No subjects will be enrolled at external national or international sites.

## 5.7 Participant Withdrawal or Termination

## 5.7.1 Reasons for Withdrawal or Termination

Participants are free to withdraw from participation in the study at any time upon request. Participation of a patient in this clinical study may be discontinued for any of the following reasons:

- The patient withdraws consent or requests discontinuation from the study for any reason;
- Occurrence of any medical condition or circumstance that exposes the patient to substantial risk and/or does not allow the patient to adhere to the requirements of the protocol;
- Any AE, clinically significant adverse event, severe laboratory abnormality, intercurrent illness, or other medical condition that indicates to the investigator that continued participation is not in the best interest of the patient;
  - Pregnancy during study period;


- Patient failure to comply with protocol requirements or study-related procedures;
  - Termination of the study by the Sponsor, the regulatory authority, FDA, or IRB.
- The participant meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation
- Progression of osteoarthritis requiring surgical therapy
- Patients found to have osteonecrosis on pre-procedural MRI

## 5.7.2 Handling of Participant Withdrawals or Termination

report form (eCRF). In the case of loss of follow-up, attempts to contact the patient will be made and documented in the patient's medical records. If a patient withdraws prematurely from the study due to the above criteria or any other reason, study staff should make every effort to complete the full panel of assessments scheduled for the follow-up visits. The reason for patient withdrawal must be documented in the electronic case Every effort will be made to undertake protocol-specified safety follow-up procedures to capture AEs, serious adverse events (SAEs), and unanticipated problems (UPs)

Withdrawn patients can be replaced.

## 5.8 Premature Termination or Suspension of Study

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to investigator, funding agency, the IDE sponsor and regulatory authorities. If the study is prematurely terminated or suspended, the PI will promptly inform the IRB and will provide the reason(s) for the termination or suspension.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable

Study may resume once concerns about safety, protocol compliance, data quality are addressed and satisfy the sponsor, IRB and/or FDA.

# Study Agent (Study device) and/or Procedural Intervention

### 6.1 Study Device Description

perfluorinated polymer (Polyzene<sup>TM</sup>-F). The microspheres intended to occlude vasculature for the purpose of blocking blood flow to a target tissue. delivery through the indicated delivery catheter and color-coded by size to allow for easy identification. 250 µm microsphere will be used and are They are available in prefilled syringes in a range of sizes suitable for embolic therapy. The microspheres are compressible to enable smooth Embozene™ Microspheres are spherical, tightly calibrated, biocompatible, nonresorbable, hydrogel microspheres coated with an inorganic supplied in prefilled yellow syringes.

hypervascular tumors, including uterine fibroids and hepatoma, and for embolization of prostatic Embozene Microspheres are intended for embolization of arteriovenous malformations and


arteries for symptomatic benign prostatic hyperplasia. This device is not intended for neurovascular use. The device is FDA approved for above indications (FDA approved for treatment of BPH; FDA approval 510(K) # K180102; 510(k) premarket notification of intent to market the device FDA 510(k) # K141209)

There are no known chemical interactions between Embozene Microspheres and pharmaceuticals.

IDE for the purpose of this study was obtained.

### 6.1.1 Acquisition

Embozene™ Microspheres will be supplied by the manufacturer.

## .1.2 Formulation, Appearance, Packaging, and Labeling

Embozene Microspheres are supplied in a 20 ml syringe prefilled with 2 ml of product suspended in a non-pyrogenic, sterile transport solution of Embozene Microspheres are packaged in a sterile, sealed tray with a peel-away lid. The label indicates the specific size of the microspheres physiological saline. The total volume of Embozene Microspheres including transport solution is approximately 7 ml. Prefilled syringes of contained in the syringe. 250 µm microsphere will be used and are supplied in prefilled yellow syringes.

## 6.1.3 Product Storage and Stability

expiration date on label. The investigational device will be stored in a secure locked cabinet in the interventional radiology storage area (Tisch As per manufacturer's instructions specified in the DFU, the device should be stored in a cool, dry, dark place. Product must be used prior to hospital,  $2^{nd}$  floor) and only the PI and research coordinator will have access to the lock.

### 6.1.4 Preparation

Embozene Microspheres are supplied in a 20 ml syringe prefilled with 2 ml of product suspended in a non-pyrogenic, sterile transport solution of physiological saline. The total volume of Embozene Microspheres including transport solution is approximately 7 ml Prior to embolization, the transport solution will be eliminated from the syringe. An embolic mixture will be prepared by adding 9 cc saline + 9 cc iodinated contrast added to the 2 cc of product (Embozene Microspheres) for a total of 20 cc embolic mixture.

### 6.1.5 Dosing and Administration

The embolic mixture will be injected in small increments until blood flow stagnates in the target artery (1 cc embolic mixture injected over 2 minutes, followed by 1 cc saline delivered slowly, then 3 cc saline flush)

### 6.1.6 Route of Administration

The embolic mixture will be injected in small increments in the target geniculate artery(ies) after selective catheterization of the target vessel(s) using a microcatheter to reach distal arteries while avoiding branches that do not feed abnormal vessels.

### 3.1.7 Duration of Therapy

Treatment will be completed during one interventional session (visit 3, day 0)


Study number: s19-00370 Version: 06.25.2024

## 3.1.8 Device Specific Considerations

Embozene microspheres are available in prefilled syringes in a range of sizes suitable for embolic therapy. 250 µm microsphere syringes will be used for this study and are supplied in prefilled yellow syringes.

## 3.2 Study Procedural Intervention(s) Description

digital subtraction angiography will be performed to depict the descending genicular artery, superior and inferior lateral genicular arteries, superior the femoral artery to maintain vascular access. Ultrasound-guided access may be used. A guiding catheter will be introduced and lower extremity technique. Femoral artery access will be obtained with a micropuncture needle set and a vascular sheath or a guiding catheter will be placed in and inferior medial genicular arteries, and the median genicular artery in all patients. Angiography will be performed to identify abnormal knee On the day of the procedure (visit 3, day 0), the subjects will be given the choice of receiving intravenous anxiolytic and analgesic medication (moderate sedation) during procedure or proceeding with local anesthetic only. Arterial access site will be prepped and draped using sterile neovasculature arising from one or more of geniculate arterial branches. After localizing the abnormal neovessels (abnormal vessels appear as tumor blush-type enhancement in the arterial phase, often accompanied by be receiving the microspheres. The abnormal vessels will be embolized with 250 µm Embozene™ Microspheres solution under direct fluoroscopic simulation can be performed with contrasted cone beam CT on the procedure table. This will allow the operators to know exactly what tissues will early venous drainage /hypervascular synovial tissue in the region of the target knee joint), a microcatheter will be inserted coaxially through the visualization to prevent reflux and non-target embolization. Multiple geniculate arteries may be embolized until neovascularity is no longer seen. guiding catheter and selectively placed in the targeted artery(ies). If there is uncertainty about the angiographic findings, pre-embolization

branches that do not feed abnormal vessels. After embolization, a repeat lower extremity angiogram and contrasted cone beam CT (if needed) will procedure. If hemostasis obtained by manual compression, it is anticipated that most participants will be discharged home 6 hours post procedure. the femoral artery sheath removal. All participants will be monitored for 2-6 hours post procedure and any adverse events will be documented and hemostasis of the arterial access will be achieved by an FDA-approved arterial closure device or manual compression and bed rest for 2-6 h after cc saline flush). In some cases, more selective catheterization will be performed by using the microcatheter to reach distal arteries while avoiding antegrade flow of contrast) in the target artery(ies) (1 cc embolic mixture injected over 2 minutes, followed by 1 cc saline delivered slowly, then 3 Injection of the embolic mixture will continue in small increments until an end point of at least 'pruning" of the hypervascular synovium ' (slowed The embolic mixture will be prepared by adding 9 cc of saline + 9 cc of contrast to the 2 cc Embosepheres for a total of 20 cc embolic mixture. managed. If hemostasis obtained by a vascular closure device, it is anticipated that most participants will be discharged home 2 hours post then be performed to evaluate for success of embolization and to exclude complication. The catheter(s) and sheath will be removed, and

Disposable syringes which spherical particulate will be discarded as medical waste and packaging will be kept in a secure location until the study is completed. Packages will be disposed of upon completion of the study.

## 6.2.1 Administration of Procedural Intervention

subject will be discharged home the same day (<23 hours) unless a complication arises that requires inpatient admission for management of the hours. Additional 2-6 hours will be needed after hemostasis of the access femoral artery is achieved for monitoring / observation. In general, the interventional procedure will be performed during one session (day 0) with an approximate duration of the procedure estimated between 1-3 Procedure will be performed by one of two interventional radiologists with fellowship training in Vascular and Interventional Radiology. The complication.


Version: 06.25.2024


## Study Procedures and Schedule

## 7.1 Study Procedures/Evaluations

### 7.1.1 Study Specific Procedures

- Medical history
- Complete medical history will be obtained from medical records if available and/or by interview during clinic visits.
- History of previous and concomitant treatment
- Knee injections and frequency over the 12 months
- Medication history over the last month will be obtained during pre and post intervention study visits. Medication history will focus on medications currently taken for the treatment of knee OA, including prescription and over-the-counter medications for pain.
  - Physical therapy and frequency over the 12 months 0
- Weight loss / gain
- Focused physical examination:
- Vital signs (temperature, blood pressure, heart rate, oxygen saturation, height, weight, BMI)
  - Focused knee examination.
- Lower extremity pulses
- Imaging assessment with knee MRI
- Baseline and follow-up (at 3 months) knee MRI will be performed.
- Knee MRI protocol will include: Axial t2 FS, Sagital PD, Sagital T2 FS, Coronal PD, Coronal PD FS, non-contrast axial and sagittal
- Imaging variables collected for this study is found in the attached eCRFs
- A discussion of the results of any study specific procedures (e.g., radiographic or other imaging or laboratory evaluations) will be provided to participant after the completion of the study unless these information represent a significant health-related issue.
- Laboratory tests:
- Baseline and follow-up (at 1-, 3-, and 12-, 18-48 months) laboratory tests will be obtained
  - Administration of questionnaires or other instruments for patient-reported outcomes:
    - Electronic VAS
- KOOS questionnaire
- Self-reported quality of life EQ-5D-5L questionnaire

## Standard of Care Study Procedures

- Standard of care imaging assessment with knee radiograph:
- Knee radiograph obtained within 6 months of the screening will be used to assess the Kellgren-Lawrence (KL score)
- A new knee radiograph will be obtained during or prior to visit 2 if no recent (within 6-month) radiograph of the target knee is available
- Knee radiograph protocol: AP weightbearing, lateral, sunrise views
- KL score will be assessed by a blinded musculoskeletal radiologist (one of co-investigators) 0 0


## 7.2 Laboratory Procedures/Evaluations

### 7.2.1 Laboratory Evaluations

Baseline laboratory tests on peripheral venous blood drown from patient during clinic visit #2 (if not available within the last 30 days prior to procedure

- Hematology: Complete blood count (CBC)
- Biochemistry: Basic metabolic panel (BMP)
- Coagulation profile: INR
- **Pregnancy test**: point pregnancy test will be performed prior to procedure as standard procedure prior to fluoroscopic examination.

Baseline and follow-up laboratory tests on urine samples and peripheral venous blood drown from patient during clinic visits (2, 5, 6, 7). Approximately 10 cc of blood will be collected from peripheral venous blood in each visit that requires collection of blood samples

- Inflammatory biomarkers:
- MMP (total activity assay),
- IL1Ra,
- sRAGE,

  - hsCRP, VEGF, 0
- S100 protein
- Pain biomarkers
- Substance P NGFb, CCL2 0
- 0
- Matrix degradation collagen biomarkers
  - CTX-II and CTX-I.
- Type IV collagen markers (C4M, PRO-C4)\*
- PRO-C6 measuring endothelium dysfunction\*
- Synovial and cartilage markers (C2M, ARGS, CRPM, C1M, C3M)\*

up to analyze multiple serum, urine, and plasma biomarkers. We are requesting IRB modification to add an optional final visit for patients who The current approved IRB protocol involves collection of blood and urine from all subjects at baseline, 1-month, 3-month, and 12-month follow completed 12 months follow up by August 31, 2024 after obtaining informed consent. This visit will include blood and urine collection similar to prior visits. No significant increase in risk. At the patient's request, this visit can be performed by a telemedicine visit, a phone call, or via a secure email to participant. In this case, the informed consent can be obtained via phone and the coordinator / investigator will sign in the presence of a If performed via email, the coordinator will send the questionnaire to patient using a secure email (sendsafe) and participants can email it back to witness. If the visit is performed via telemedicine or phone call, the research coordinator will ask the patient the questions and document the answers.


of having a longer follow up with study team. If the visit is performed remotely, blood and urine samples, used for biomarkers and exploratory analysis research coordinator or PI. This addition of a virtual visit will not increase the risk of participants; in contrary, it will provide the patient with the benefit points, will not be required.

to outside laboratory /subcontractors. These additional biomarkers are marked with an Asterix above are: type IV collagen markers (C4M, PRO-\* A portion of the collected material as part of the approved protocol, including blood, and urine, may be sent for additional biomarker analysis C4); PRO-C6 measuring endothelium dysfunction; synovial and cartilage markers (C2M, ARGS, CRPM, C1M, C3M). All samples sent to outside collaborations / laboratories will be deidentified by date of collection and barcode as identifiers to protect subjects' identity. No additional samples will be collected as part of the modification. No additional risks to subjects are expected.

- Optional segment: The evaluation of the ADDITIONAL biomarkers in the outside lab will be optional for subjects. The biomarker analysis performed by IR-approved study team members at NYU will remain unchanged as part of the modification.
- identified by barcodes and collection date only and kept in the NYU Langone Orthopedic Hospital. When samples are sent to an outside Storage location: These samples (serum, plasma, and urine samples collected as part of the approved research protocol are stored and aboratory (optional part of the study), the remaining samples will be discarded after the biomarker analysis is performed and results obtained.
- Access to samples: IRB-approved study team members from NYU Langone Orthopedic Hospital have access to these samples.
- Protecting subject anonymity: Study team members who have access to the samples will received the blood / urine tubes labeled with study subject number and date of collection.
- Samples will be stored until the end of data analysis and study closure. All samples sent to outside collaborations / laboratories will be de-identified by date of collection and barcode

### 7.3 Study Schedule

### 7.3.1 Screening

# Screening Visit (Visit 1, Day -30 to -2)- In rheumatology or vascular and interventional radiology clinic

- Obtain informed consent of potential subject (If the subject wishes to take more time to review the study before enrolling, he/she may complete the consent process at the beginning of the next visit)
- Provide a copy of informed consent and study brochure to subject
- Review subject's eligibility based on inclusion/exclusion criteria
- Collect demographic variables
  - Obtain medical history
- Schedule study visits for eligible participants


Note: if subject prefers, visits 1 and 2 can be combined and procedures of these visits may be performed on the same day after screening and obtaining informed consent.


Those candidates who are disqualified from study entry will be logged into the Screening Log with a reason for no study entry. A copy of the consent will be provided to the subject and the original filed in the study files.

## Enrollment/Baseline (Visit 2, Day -29 to -1)- In interventional radiology clinic 7.3.2

- Verify informed consent of potential participant (study consent)
- Verify subject's eligibility
- Targeted physical exam
- Administration of study questionnaires
- Previous / concomitant treatments
- Baseline MRI (if one is not available within the last 3 months)
- Baseline knee radiograph (if one is not available within the last 6 months)
- Peripheral venous blood draws and urine sample (baseline laboratory tests)
- Note: Subjects will be required to withhold pain medications 24 hours prior to screening and each visit for the evaluation of pain

## 7.3.3 Interventional visit (visit 3, Day 0)

- Within 30 days of visit 1
- Verify informed consent of participant verified by signature on written informed consent
- Geniculate artery embolization
- Record any immediate complications / adverse events detected during the procedure or observation period (if applicable)
- Subjects will be given a phone number to reach a physician 24 hours a day to report any adverse symptoms and receive medical advice

### 7.3.4 Follow-up Visits

## 7.3.4.1 Follow up visit at 1 day (Visit #4; day 1 /+3 days)

Subjects will be seen in clinic or contacted by phone or per the subject's preference the day following GAE (+3 days). As most complications of the procedure will be evident within this time period, this visit is to evaluate for early AE's. If AE is suspected based on change in pain scores or functionality, further assessment and management will be performed based on the nature of suspected adverse event.

## 7.3.4.2 Follow up visit at 1-month (Visit 5, Day 30 +/- 10)

- Obtain medical history
- Record adverse events as reported by participant or observed by investigator (if applicable)
- Targeted physical exam
- Administration of study questionnaires
- Previous / concomitant treatments, including medical history
- Peripheral venous blood draw and urine sample to perform follow-up laboratory tests


Note: Subjects will be required to withhold pain medications 24 hours prior to screening and each visit for the evaluation of pain

## 7.3.4.3 Follow up visit at 3 months (Visit 6, Day 90 +/- 10)

- Obtain medical history
- Record adverse events as reported by participant or observed by investigator (if applicable)
- Targeted physical exam
- Administration of study questionnaires
- Previous / concomitant treatments, including medical history
- Peripheral venous blood draw and urine sample to perform follow-up laboratory tests
- Follow-up knee MRI
- Note: Subjects will be required to withhold pain medications 24 hours prior to screening and each visit for the evaluation of pain

## 7.3.4.4 Follow up visit at 12 months (Visit 7, Day 360 +/- 10)

- Obtain medical history
- Record adverse events as reported by participant or observed by investigator (if applicable)
- Targeted physical exam
- Administration of study questionnaires
- Previous / concomitant treatments, including medical history
- Peripheral venous blood draw and urine sample to perform follow-up laboratory tests
- Note: Subjects will be required to withhold pain medications 24 hours prior to screening and each visit for the evaluation of pain

## 7.3.5 Follow up visit at 18-48 month (visit 8):

- This visit is optional to all study participants who completed 12 months visit by August 31, 2024 and fall within 18-48 months window from the date of procedure. This visit is not expected to add significant risk to participant and will only occur after obtaining informed consent from participants. This visit is important to add at this point of the trial to obtain long term follow up data.
- Obtain medical history
- Record adverse events as reported by participant or observed by investigator (if applicable)
- Targeted physical exam
- Administration of study questionnaires
- Previous / concomitant treatments, including medical history
- Peripheral venous blood draw and urine sample to perform follow-up laboratory tests
- Note: Subjects will be required to withhold pain medications 24 hours prior to screening and each visit for the evaluation of pain

## 7.3.6 Withdrawal/Early Termination Visit

- Obtain medical history
- Record adverse events as reported by participant or observed by investigator (if applicable)
- Targeted physical exam


Version: 06.25.2024

- Administration of study questionnaires
- Previous / concomitant treatments, including medical history
- Peripheral venous blood draw and urine sample to perform follow-up laboratory tests
- Note: Subjects will be required to withhold pain medications 24 hours prior to screening and each visit for the evaluation of pain

### 7.3.7 Unscheduled Visit

Unscheduled visits if needed will be documented in the medical chart of the subject including the reason for the visit and assessment / management plan as determined by the visit.

## 7.4 Concomitant Medications, Treatments, and Procedures

Medications to be reported in the eCRF are concomitant prescription medications, over-the-counter medications and non-prescription medications used pain management. For this protocol, a prescription medication is defined as a medication that can be prescribed only by a properly All relevant concomitant medications taken during study participation, as well as treatments and procedures will be recorded on eCRFs. authorized/licensed clinician.

Note: Subjects will be required to withhold pain medications 24 hours prior to screening and each visit for the evaluation of pain

## Rescue Medications, Treatments, and Procedures

In the event of non-target embolization during the procedural visit leading to limb ischemia, subsequent interventions and / or medical management may be required for treatment of limb ischemia.

## Participant Access to Study Agent at Study Closure

After participants are no longer enrolled in the study, they will return to standard of care treatment for knee OA.

### **Assessment of Safety** $\infty$

## Specification of Safety Parameters

Safety parameters include the number, severity, causality, timing, and description of complications, adverse events, or poor outcomes that are secondary to the procedure.
Version: 06.25.2024

## 8.1.1 Definition of Adverse Events (AE)

Intercurrent illnesses or injuries should be regarded as adverse events. Abnormal results of diagnostic procedures on target knee in the follow-up period after the study intervention are considered to be adverse events if the abnormality: An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study

- results in study withdrawal
- is associated with a serious adverse event
- is associated with clinical signs or symptoms
- leads to additional treatment or to further diagnostic tests
- is considered by the investigator to be of clinical significance

### Definition of Serious Adverse Events (SAE) 8.1.2

Serious adverse events are considered to be those resulting in an unplanned increase in the level of care, prolonged hospitalization, permanent adverse sequelae, or death

## A serious adverse event is any AE that is:

- life- or limb- threatening
- requires or prolongs hospital stay
- results in persistent or significant disability or incapacity
- a congenital anomaly or birth defect
- an important medical event

Important medical events are those that may not be immediately life or limb threatening but are clearly of major clinical significance. They may eopardize the subject and may require intervention to prevent one of the other serious outcomes noted above.

All adverse events that do not meet any of the criteria for serious should be regarded as non-serious adverse events.

# Definition of Unanticipated Problems (UP)

Unanticipated Problems Involving Risk to Subjects or Others

Any incident, experience, or outcome that meets all of the following criteria:

- Unexpected in nature, severity, or frequency (i.e. not described in study-related documents such as the IRB-approved protocol or consent form, the investigators brochure, etc)
- Related or possibly related to participation in the research (i.e. possibly related means there is a reasonable possibility that the incident experience, or outcome may have been caused by the procedures involved in the research)
- Suggests that the research places subjects or others at greater risk of harm (including physical, psychological, economic, or social harm).


investigational plan or application, or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare Unanticipated adverse device effect, any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the of subjects (21 CFR 812.3(s))

## 8.2 Classification of an Adverse Event

### 8.2.1 Severity of Event

severe, life-threatening / disabling event, or death/ unexpected pregnancy abortion. The investigator will also categorize each adverse event as to The Investigator will assess the severity (intensity) of each adverse event as mild, moderate, ts potential relationship to study drug using the categories of yes or no.

The severity and causality of all adverse events will be graded according to the new adverse event classification by the Society of Interventional Radiology Standards of Practice Committee [30], as follows:

- Mild AE: No therapy or nominal (non-substantial) therapy (postprocedural imaging performed and fails to show manifestation of AE); near miss (eg, wrong site of patient prepared, recognized and corrected before procedure, wrong patient information entered for procedure);
  - intervention) under conscious sedation, blood product administration, extremely prolonged outpatient observation, or overnight admission **Moderate AE:** moderate escalation of care, requiring substantial treatment, eg, intervention (description of intervention and result of after outpatient procedure not typical for the procedure (excludes admission or hospital days unrelated to AE);
    - general anesthesia would primarily be used in lieu of conscious sedation, eg, in mentally challenged or severely uncooperative patients); admission that is atypical for the procedure, inpatient transfer from regular floor/telemetry to intensive care unit, or complex intervention performed requiring general anesthesia in previously non-intubated patient (generally excludes pediatrics or in circumstances in which Severe AE: marked escalation of care, ie, hospital admission or prolongation of existing hospital admission for > 24 hours, hospital
      - Life-threatening or disabling event: eg, cardiopulmonary arrest, shock, organ failure, unanticipated dialysis, paralysis, loss of limb or
        - Patient death or unexpected pregnancy abortion.

For AEs not included in the protocol defined grading system, the following guidelines will be used to describe severity.

- **Mild** Events require minimal or no treatment and do not interfere with the participant's daily activities.
- Moderate Events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
- Severe Events interrupt a participant's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating.

## 8.2.2 Relationship to Study Device

For all collected AEs, the clinician who examines and evaluates the participant will determine the AE's causality based on temporal relationship and his/her clinical judgment. The degree of certainty about causality will be graded using the categories below according to the new adverse event classification by the Society of Interventional Radiology Standards of Practice Committee

- Category 1: AE not caused by procedure. The AE is completely independent of study drug administration, and/or evidence exists that the event is definitely related to another etiology. There must be an alternative, definitive etiology documented by the clinician.
- Category 2: Unknown whether AE was caused by the procedure.
- Category 3: AE caused by the procedure. There is clear evidence to suggest a causal relationship, and other possible contributing factors

study device. This means that there are facts (evidence) or arguments to suggest a causal relationship. The definition implies a reasonable possibility of a causal relationship between the event and the

The following factors should also be considered:

- The temporal sequence from study procedure: The event should occur after the study procedure. The length of time from study procedure to event should be evaluated in the clinical context of the event.
- Underlying, concomitant, intercurrent diseases: Each report should be evaluated in the context of the natural history and course of the disease being treated and any other disease the patient may have.
- Concomitant procedures / treatments: The other drugs the patient is taking or the treatment the patient receives should be examined to determine whether any of them might be recognized to cause the event in question.
- Known response pattern for this class of study procedure: Clinical and/or nonclinical data may indicate whether a particular response is likely to be a class effect.
- Exposure to physical and/or mental stresses: The exposure to stress might induce adverse changes in the recipient and provide a logical and better explanation for the event.

### 8.2.3 Expectedness

The PI will be responsible for determining whether an AE is expected or unexpected. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study device.

# Time Period and Frequency for Event Assessment and Follow-Up

relationship to study procedure (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of The occurrence of an AE or SAE may come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by one of investigators. All AEs including local and systemic reactions not meeting the criteria for SAEs will be the event. All AEs occurring while on study must be documented appropriately regardless of relationship. All AEs will be followed to adequate captured on the appropriate eCRF. Information to be collected includes event description, time of onset, clinician's assessment of severity, resolution

However, if the study participant's condition deteriorates at any time during the study, it will be recorded as an AE. UPs will be recorded in the data Any medical condition that is present at the time that the participant is screened will be considered as baseline and not reported as an AE. collection system throughout the study.


Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

days (for SAEs) after the last day of study participation. At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the The PI will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 last visit. Events will be followed for outcome information until resolution or stabilization.

reasonably be related to this study. The sponsor should also be notified if the investigator should become aware of the development of cancer or All unresolved adverse events should be followed by the investigator until the events are resolved, the subject is lost to follow-up, or the adverse subject, or the subject's personal physician, believes might reasonably be related to participation in this study. The investigator should notify the event is otherwise explained. At the last scheduled visit, the investigator should instruct each subject to report any subsequent event(s) that the study sponsor of any death or adverse event occurring at any time after a subject has discontinued or terminated study participation that may of a congenital anomaly in a subsequently conceived offspring of a subject that has participated in this study.

# 8.4 Reporting Procedures – Notifying the IRB

## 8.4.1 Adverse Event Reporting

The principal investigator will promptly notify the IRB of any unanticipated problems involving risks to subjects or others that occurs during the course of a study within five working days of learning about the event using Research Navigator.

## 3.4.2 Serious Adverse Event Reporting

principal investigator will promptly notify the IRB of any unanticipated problems involving risks to subjects or others that occurs during the course Serious adverse events will be captured from the time of the main study's informed consent through 30 days after the last follow-up visit. The of a study within five working days of learning about the event using Research Navigator.

The investigators shall submit to the sponsor and to the reviewing IRB a report of any unanticipated adverse device effect occurring during an investigation as soon as possible, but in no event later than 10 working days after the investigator first learns of the effect.

FDA and to all reviewing IRB's and participating investigators within 10 working days after the sponsor first receives notice of the effect. Thereafter The sponsors who conducts an evaluation of an unanticipated adverse device effect under 812.46(b) shall report the results of such evaluation to the sponsor shall submit such additional reports concerning the effect as FDA requests

## 8.4.3 Unanticipated Problem Reporting

Incidents or events that meet the OHRP criteria for UPs require the creation and completion of an UP report form. It is the site investigator's responsibility to report UPs to their IRB and to the DCC/study sponsor. The UP report will include the following information:

- Protocol identifying information: protocol title and number, PI's name, and the IRB project number;
  - A detailed description of the event, incident, experience, or outcome;


- An explanation of the basis for determining that the event, incident, experience, or outcome represents an UP;
- A description of any changes to the protocol or other corrective actions that have been taken or are proposed in response to the UP.

To satisfy the requirement for prompt reporting, UPs will be reported using the following timeline:

- UPs that are SAEs will be reported to the IRB and to the DCC/study sponsor within 5 working days of the investigator becoming aware of the event
- Any other UP will be reported to the IRB and to the DCC/study sponsor within 10 working days of the investigator becoming aware of the problem.

### Reporting of Pregnancy 8.4.4

If the subject participating in the study is found to be pregnant during the study period, participant will immediately be withdrawn from the study and IRB will be informed.

## Reporting Procedures – Notifying the Study Sponsor 8.5

The study clinician will complete a SAE Form within the following timelines:

- All deaths and immediately life-threatening events, whether related or unrelated, will be recorded on the SAE Form and submitted to the study sponsor (PI) within 24 hours of awareness.
- Other SAEs regardless of relationship will be submitted to the study sponsor (PI) within 72 hours of site awareness.

All SAEs will be followed until satisfactory resolution or until the site investigator deems the event to be chronic or stable. Other supporting documentation of the event may be requested by the study sponsor and should be provided as soon as possible.

applicable, on the unanticipated event or the unanticipated problem in the form of a written narrative. This should include a copy of the completed Unanticipated Problem form, and any other diagnostic information that will assist the understanding of the event. Significant new information on As a follow-up to the initial report, within the following 48 hours of awareness of the event, the investigator shall provide further information, as ongoing unanticipated adverse effects shall be provided promptly to the study sponsor.

## Reporting Procedures – Notifying the FDA 8.6

The study sponsor is required to report certain study events in an expedited fashion to the FDA. These written notifications of adverse events are referred to as IDE safety reports

- Within 10 working days (via telephone or facsimile report) Any study event that is:
  - associated with the use of the study device, and
    - unanticipated

regardless of the seriousness of the event.


Within 5 working days (via written report)

- Protocol deviation to protect the life of the subject in emergency
  - Withdrawal of IRB approval
- Lack of informed consent

## Additional reporting requirements

Sponsors are also required to identify in IDE safety reports all previous reports concerning similar adverse events and to analyze the significance of the current event in light of the previous reports.

### Reporting Process

Adverse events may be submitted on FDA Form 3500A (MEDWATCH Form) [attachment 9], or in a narrative format.

## 8.7 Safety Oversight

appropriate reporting of adverse events as noted above, as well as the construction and implementation of a site data and safety-monitoring plan. Medical monitoring will include a regular assessment of the number and type of serious adverse events. Data (demographics, eligibility criteria), It is the responsibility of the Principal Investigator to oversee the safety of the study. This safety monitoring will include careful assessment and screening methods, and adverse events will be assessed by the PI who is a fellowship trained interventional radiologist and licensed physician monthly to ensure study safety, compliance, and integrity/accuracy of data in accordance with the data safety monitoring plan.

(PI). The PI will notify the study investigators immediately when the third grade 3 event is reported and enrollment screens will stop accepting new Administration of study procedure will be halted when three moderate or higher grade AEs determined to be "related" are reported to the sponsor provide recommendations for proceeding with the study. The study sponsor will inform the IRB and FDA of the temporary halt and the disposition study participants. The study sponsor will convene a meeting with study investigators by teleconference or in writing as soon as possible and will

The outcomes of these reviews, when adverse events are captured will be communicated directly with the IRB. A summary of these reviews will be submitted to the IRB as part of an annual progress report at Continuing Review.

Specific data safety monitoring plan is listed below:

- 1- Vascular injury / non-target embolization to lower extremity, bleeding, access site complications will be monitored as follows:
- On the day of procedure, interventional radiologist (investigator) performing the procedure will assess access site and lower extremity pulses and document
- Day 1 visit / telemedicine visit: investigator will assess for symptoms in the target lower extremity (pain, swelling at access site and document findings <u>ە</u>
  - 4 weeks follow up visit: investigator will assess groin access site for hematoma, pseudoaneurysm and assess lower extremity bulses ပ
- Skin ulceration, cutaneous purpura, plantar or peripheral sensory paresthesia will be monitored as follows:
- Each follow up visit, an investigator will assess for symptoms and signs in the target lower extremity and document


# 9 Clinical Monitoring/Quality Assurance

accurate, complete, and verifiable, and that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, Clinical site monitoring is conducted to ensure that the rights and well-being of human subjects are protected, that the reported trial data are and with applicable regulatory requirement(s).

- Monitoring for this study will be performed by the study PI once every 3 months.
- Monitoring activities include communication with the sub-investigators and study site staff; review of the study site's processes, procedures, and records; and verification of the accuracy of data.

## 10 Statistical Considerations

# 10.1 Statistical and Analytical Plans (SAP)

A formal SAP will not be performed prior to database lock since this study is a pilot study with no randomization.

## 10.2 Statistical Hypotheses

assessment of whether or not each patient shows at least a 50% reduction in WOMAC pain scores from baseline (pre-treatment) to post-treatment This is a single arm study (i.e., no sham, placebo or alternative treatment included). The primary objective (clinical success rate) is a binary follow-up at 3 months. The study is designed to test the null hypothesis (H0) that the true proportion (PT) of patients that will manifest a positive treatment response, is no greater than 0.5 against the one-sided alternative hypothesis (HA) that PT ≥ 0.75. The null hypothesis will be rejected and it will be concluded that the treatment is worthy of further investigation if at least 16 of the 23 patients show a positive response to treatment.

The response rate will be summarized in terms of the observed proportion of patients manifesting a positive response and a two-sided exact 95% confidence interval (CI) per the Blyth-Still-Casella method (31). The treatment will be declared a success if the data support the conclusion that at least 75% of treated patients can be expected to show a positive response. The treatment will be considered unworthy of additional study without further development if the data are consistent with the conclusion that no more than 50% of treated patients can be expected to show a positive response.

## 10.3 Analysis Datasets

Participants who complete all follow-up visits will be included in the study.

Study number: s19-00370 Version: 06.25.2024

## 10.4 Description of Statistical Methods

The response rate will be summarized in terms of the observed proportion of patients manifesting a positive response and a two-sided exact 95% confidence interval (CI) per the Blyth-Still-Casella method (31).

## 10.4.1 General Approach

be summarized in terms of the observed proportion of patients manifesting a positive response and a two-sided exact 95% confidence interval (CI) treatment follow-up at 3 months without an increase in baseline incidence of pain medication use or intra-articular injection. The response rate will as a binary outcome of whether or not each patient shows at least a 50% reduction in WOMAC pain scores from baseline (pre-treatment) to post-This is a single arm study (i.e., no sham, placebo or alternative treatment included). The primary objective (clinical success rate) will be assessed per the Blyth-Still-Casella method. WOMAC pain score, pain VAS, WOMAC stiffness and physical activity scores will be assessed as mean and standard deviation.

## 10.4.2 Analysis of the Primary Endpoint(s)

The primary endpoint is the clinical success rate defined as at least 50% reduction in WOMAC pain score at 3-month follow-up compared to baseline as a binary assessment.

# 10.4.3 Analysis of the Secondary Endpoint(s)

or any adverse event); (4) reduction in the usage of pain medication, the frequency of infection therapy, the need for physical therapy; and (5) the treatment follow-up visit. Changes in the outcomes from baseline to follow-up will be tested using the paired-sample Wilcoxon signed rank test for function scores and the total WOMAC knee physical function score; (2) the technical success rate (defined as the proportion of patients for whom Analysis of secondary endpoints include: (1) changes in the mean WOMAC and VAS pain scores, the mean WOMAC knee stiffness and physical the procedure was successfully completed); (3) the adverse event rate (defined as the proportion of patients showing each type of adverse event the WOMAC and VAS scores and the McNemar test for the other measures which will be assessed as binary outcomes (e.g., whether or not the proportion of patients showing synovial thickening, joint effusion, meniscus tear, synovial enhancement, osteophytes. A point estimate and 95% confidence interval will be provided for each secondary outcome at each time and for the change in each outcome from baseline to each postpatient reported usage of pain medication on a daily basis).

### 10.4.4 Safety Analyses

Safety endpoints will assess adverse event rate (defined as the proportion of patients showing each type of adverse event or any adverse event). The severity and causality of all adverse events will be graded according to the new adverse event classification by the Society of Interventional Radiology Standards of Practice Committee [30]

### 10.5 Sample Size

The sample size was initially selected based on primary objective so that the study will have 80% power at the 5% significance level for testing the positive treatment response. As a result, the study will accrue 23 patients since this sample size will endow the test with 80.4% power at a realized significance level of 0.047. with 20% attrition, the study will need 29 patients. We are requesting increase in the sample size to 40. With 20% with 20% attrition, the study will need to enroll 50 patients. The PI and sub-investigators determined that increase in the sample size is necessary to null hypothesis H0. PT ≤ 0.5 against the alternative hypothesis HA. PT ≥ 0.75, where PT is the true proportion of patients that will manifest a


collecting samples for biomarker analysis and the need for a larger sample size to evaluate changes in biomarker levels, an increase in sample evaluate the role of GAE as a disease-modifying treatment option for knee OA. Since this current study is the only active study in the U.S size is needed.

# 11 Source Documents and Access to Source Data/Documents

Source data is all information, original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction hospital records, clinical and office charts, laboratory notes, memoranda, subjects' diaries or evaluation checklists, pharmacy dispensing records, photographic negatives, microfilm or magnetic media, x-rays, subject files, and records kept at the pharmacy, at the laboratories, and at medicotechnical departments involved in the clinical trial. It is acceptable to use CRFs as source documents. Data collected on electronic CRFs using and evaluation of the trial. Source data are contained in source documents. Examples of these original documents, and data records include: recorded data from automated instruments, copies or transcriptions certified after verification as being accurate and complete, microfiches, TrialMaster are attached to this protocol (see attachment 4).

"N/D". If the item is not applicable to the individual case, write "N/A". All entries should be printed legibly in black ink. If any entry error has been made, to correct such an error, draw a single straight line through the incorrect entry and enter the correct data above it. All such changes must be initialed and dated. DO NOT ERASE OR WHITE OUT ERRORS. For clarification of illegible or uncertain entries, print the clarification above missing data must be explained. If a space on the CRF is left blank because the procedure was not done or the question was not asked, write The study case report form (CRF) is the primary data collection instrument for the study. All data requested on the CRF must be recorded. All the item, then initial and date it.

and inspections by the IRB/EC, the sponsor, government regulatory bodies, and University compliance and quality assurance groups of all study Access to study records will be limited to IRB-approved members of the study team. The investigator will permit study-related monitoring, audits, related documents (e.g. source documents, regulatory documents, data collection instruments, study data etc.). The investigator will ensure the capability for inspections of applicable study-related facilities (e.g. pharmacy, diagnostic laboratory, etc.).

Participation as an investigator in this study implies acceptance of potential inspection by government regulatory authorities and applicable University compliance and quality assurance offices.

# 12 Quality Assurance and Quality Control

QC procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated for clarification/resolution. The PI will verify that the clinical trial is conducted and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirements (e.g., Good Laboratory Practices (GLP), Good Manufacturing Practices (GMP))

The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.


# 13 Ethics/Protection of Human Subjects

### 13.1 Ethical Standard

All investigators will ensure that this study is conducted in full conformity with Regulations for the Protection of Human Subjects of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and/or the ICH E6.

## 13.2 Institutional Review Board

Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the IRB for review and approval. review and approval by the IRB before the changes are implemented to the study. All changes to the consent form will be IRB approved; a determination will be made regarding whether previously consented participants need to be re-consented.

## 13.3 Informed Consent Process

# 13.3.1 Consent/Assent and Other Informational Documents Provided to Participants

Consent forms describing in detail the study agent, study procedures, and risks are given to the participant and written documentation of informed consent is required prior to starting intervention/administering study product. The consent form is submitted with this protocol (See attachment 9).

# 13.3.2 Consent Procedures and Documentation

the study with their surrogates or think about it prior to agreeing to participate. The participant will sign the informed consent document prior to any the signed informed consent document will be given to the participants for their records. The rights and welfare of the participants will be protected opportunity to carefully review the written consent form and ask questions prior to signing. The participants should have the opportunity to discuss Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participants. Participants will have the Consent forms will be IRB approved and the participant will be asked to read and review the document. The investigator will explain the research procedures being done specifically for the study. The participants may withdraw consent at any time throughout the course of the trial. A copy of study participation. Extensive discussion of risks and possible benefits of participation will be provided to the participants and their families study to the participant and answer any questions that may arise. All participants will receive a verbal explanation in terms suited to their by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

individual obtaining consent, will be thoroughly documented in the subject's research record. Any alteration to the standard consent process (e.g. A copy of the signed informed consent document will be stored in the subject's research record. The consent process, including the name of the use of a translator, consent from a legally authorized representative, consent document presented orally, etc.) and the justification for such alteration will likewise be documented.

# 13.4 Participant and Data Confidentiality

Information about study subjects will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed subject authorization informing the subject of the following

- What protected health information (PHI) will be collected from subjects in this study
- Who will have access to that information and why
  - Who will use or disclose that information
- The rights of a research subject to revoke their authorization for use of their PHI.

collected prior to the revocation of subject authorization. For subjects that have revoked authorization to collect or use PHI, attempts should be In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information made to obtain permission to collect at least vital status (i.e. that the subject is alive) at the end of their scheduled study period

Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their agents. This the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

product may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, The study monitor, other authorized representatives of the sponsor, representatives of the IRB or pharmaceutical company supplying study clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by local IRB and Institutional regulations.

Langone Health. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will research staff will be the Institution-approved, encrypted and HIPAA-compliant version of TrialMastermanaged by MCIT. At the end of the study, Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at NYU be identified by a unique study identification number. The study data entry and study management systems used by NYU Langone Health all study databases will be de-identified and archived at the NYU Langone Health.

# 13.4.1 Research Use of Stored Human Samples, Specimens, or Data

- Intended Use: data collected under this protocol may be used to study knee OA. No genetic testing will be performed.
- study. . Data will be stored only on Trail Master and electronic medical records (EPIC). Data will be kept in password-protected computers. Storage: Access to stored samples will be limited to study personnel. Samples will be destroyed after the termination or completion of the Only investigators will have access to the data.

## 13.5 Future Use of Stored Specimens

Biospecimens collected for the study will not be stored for future research beyond the scope of the study


# 14 Data Handling and Record Keeping

# 14.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site PI. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

clarity of reproduced copies. When making changes or corrections, cross out the original entry with a single line, and initial and date the change. DO NOT ERASE, OVERWRITE, OR USE CORRECTION FLUID OR TAPE ON THE ORIGINAL. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data. Black ink is required to ensure

Copies of the electronic CRF (eCRF) will be provided for use as source documents and maintained for recording data for each participant enrolled in the study. Data reported in the eCRF derived from source documents should be consistent with the source documents or the discrepancies should be explained and captured in a progress note and maintained in the participant's official electronic study record.

Clinical data (including AEs, concomitant medications, and expected adverse reactions data) and clinical laboratory data will be entered into Trial Master internal, a 21 CFR Part 11-compliant data capture system provided by NYU Langone. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be entered directly from the source documents.

## 14.2 Study Records Retention

Study documents will be retained for the longer of 3 years after close-out, 5 years after final reporting/publication, or 2 years after the last approval discontinued and FDA is notified if no application is to be filed or if the application has not been approved for such indication. No records will be destroyed without the written consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the investigator when these of a marketing application is approved for the device for the indication for which it is being investigated or 2 years after the investigation is documents no longer need to be retained.

## 14.3 Protocol Deviations

may be either on the part of the participant, the investigator, or the study site staff. As a result of deviations, corrective actions are to be developed A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or Manual of Procedures (MOP) requirements. The noncompliance by the site and implemented promptly.

These practices are consistent with ICH E6:

- 4.5 Compliance with Protocol, sections 4.5.1, 4.5.2, and 4.5.3
- 5.1 Quality Assurance and Quality Control, section 5.1.1
  - 5.20 Noncompliance, sections 5.20.1, and 5.20.2.

It is the responsibility of the site PI/study staff to use continuous vigilance to identify and report deviations within 10 working days of identification of the protocol deviation, or within 10 working days of the scheduled protocol-required activity

All protocol deviations must be addressed in study source documents, reported to PI, IRB, and FDA


Protocol deviations must be reported to the local IRB per their guidelines. The site PI/study staff is responsible for knowing and adhering to their IRB requirements. Further details about the handling of protocol deviations will be included in the MOP.

## 14.4 Publication and Data Sharing Policy

ICMJE policy, and the Section 801 of the Food and Drug Administration Amendments Act of 2007, requires that all clinical trials be registered in a The ICMJE does not review specific studies to determine whether registration is necessary; instead, the committee recommends that researchers nterventions include drugs, surgical procedures, devices, behavioral treatments, process-of-care changes, and the like. Health outcomes include public trials registry such as ClinicalTrials.gov, which is sponsored by the National Library of Medicine. Other biomedical journals are considering for publication. The ICMJE defines a clinical trial as any research project that prospectively assigns human subjects to intervention or concurrent The International Committee of Medical Journal Editors (ICMJE) member journals have adopted a clinical trials registration policy as a condition responsibility to register the trial in an acceptable registry, so the research results may be considered for publication in ICMJE member journals. any biomedical or health-related measures obtained in patients or participants, including pharmacokinetic measures and adverse events. The who have questions about the need to register err on the side of registration or consult the editorial office of the journal in which they wish to adopting similar policies. For interventional clinical trials performed under NIH IC grants and cooperative agreements, it is the grantee's comparison or control groups to study the cause-and-effect relationship between a medical intervention and a health outcome. Medical

FDAAA mandates that a "responsible party" (i.e., the sponsor or designated principal investigator) register and report results of certain "applicable clinical trials":

- Trials of Drugs and Biologics: Controlled, clinical investigations, other than Phase I investigations of a product subject to FDA regulation;
- Trials of Devices: Controlled trials with health outcomes of a product subject to FDA regulation (other than small feasibility studies) and pediatric postmarket surveillance studies.

### 15 Study Finances

### 15.1 Funding Source

Varian Medical Systems, Inc are providing the device

## 15.2 Costs to the Participant

There will be no cost to participants.


# 15.3 Participant Reimbursements or Payments

No reimbursement or payments will be offered to participate in this study.

## 16 Study Administration

## 16.1 Study Leadership

The Steering Committee will govern the conduct of the study. The Steering Committee will be composed of the PI and a study co-investigator (A. Sista, MD).

## 17 Conflict of Interest Policy

appropriate to their participation in the trial. The study leadership has established policies and procedures for all study group members to disclose The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore any actual managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest. Any investigator who has a conflict of interest with this study (patent ownership, royalties, or financial gain greater than the minimum allowable by sanctioned conflict management plan that has been reviewed and approved by the study sponsor prior to participation in this study. All NYULMC their institution, etc.) must have the conflict reviewed by the NYU Langone Conflict of Interest Management Unit (CIMU) with a Committeeinvestigators will follow the applicable conflict of interest policies.

### 18 References

- Bijlsma JW, Berenbaum F, Lafeber FP: Osteoarthritis: an update with relevance for clinical practice. Lancet 2011, 377:2115-2126. <del>1.</del> 4.
  - Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, et al: The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis 2014, 73:1323-1330.
    - Peat G, McCarney R, Croft P: Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Annals of the rheumatic diseases 2001, 60:91-97 ω.
- Blagolevic M, Jinks C, Jeffery A, Jordan KP: Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage 2010, 18:24-33. 4.
  - Litwic A, Edwards MH, Dennison EM, Cooper C: Epidemiology and burden of osteoarthritis. Br Med Bull 2013, 105:185-199. 6.5
- Okuno Y, Korchi AM, Shinjo T, Kato S: Transcatheter arterial embolization as a treatment for medial knee pain in patients with mild to moderate osteoarthritis. Cardiovascular and interventional radiology 2015, 38:336-343.
  - McAlindon TE, Bannuru RR, Sullivan M, Arden N, Berenbaum F, Bierma-Zeinstra S, Hawker G, Henrotin Y, Hunter D, Kawaguchi H: OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis and cartilage 2014, 22:363-388. ۲.


effectiveness, practice variations, indications and possible determinants of utilization. Rheumatology (Oxford) 1999, 38:73-83. Dieppe P, Basler HD, Chard J, Croft P, Dixon J, Hurley M, Lohmander S, Raspe H: Knee replacement surgery for osteoarthritis:

- Dieppe P, Lim K, Lohmander S: Who should have knee joint replacement surgery for osteoarthritis? International journal of rheumatic diseases 2011, 14:175-180. <u>ග</u>
- Mapp PI, Walsh DA: **Mechanisms and targets of angiogenesis and nerve growth in osteoarthritis.** N*ature Reviews Rheumatology* 6.
- Ashraf S, Mapp PI, Walsh DA: Contributions of angiogenesis to inflammation, joint damage, and pain in a rat model of osteoarthritis. Arthritis & Rheumatism 2011, 63:2700-2710. 7
- Ashraf S, Wibberley H, Mapp PI, Hill R, Wilson D, Walsh DA: Increased vascular penetration and nerve growth in the meniscus: a potential source of pain in osteoarthritis. Annals of the rheumatic diseases 2011, 70:523-529. 12
  - Mapp P, Avery P, McWilliams D, Bowyer J, Day C, Moores S, Webster R, Walsh D: **Angiogenesis in two animal models of** osteoarthritis. Osteoarthritis and cartilage 2008, 16:61-69. <del>1</del>3
- Suri S, Gill SE, de Camin SM, McWilliams DF, Wilson D, Walsh DA: Neurovascular invasion at the osteochondral junction and in osteophytes in osteoarthritis. Annals of the rheumatic diseases 2007, 66:1423-1428. 4.
- Walsh D, Bonnet C, Turner E, Wilson D, Situ M, McWilliams D: Angiogenesis in the synovium and at the osteochondral junction in osteoarthritis. Osteoarthritis and cartilage 2007, 15:743-751. 15.
- measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW: Validation study of WOMAC: a health status instrument for or knee. The Journal of rheumatology 1988, 15:1833-1840. 16.
  - Peterfy C, Guermazi A, Zaim S, Tirman P, Miaux Y, White D, Kothari M, Lu Y, Fye K, Zhao S: Whole-organ magnetic resonance imaging score (WORMS) of the knee in osteoarthritis. Osteoarthritis and Carilage 2004, 12:177-190 17.
- recanalization of four different spherical embolization agents in the porcine kidney model. Journal of Vascular and Interventional Stampfl S, Bellemann N, Stampfl U, Radeleff B, Lopez-Benitez R, Sommer C-M, Thierjung H, Berger I, Richter GM: Inflammation and Radiology 2008, 19:577-586. <del>0</del>
- Biocompatibility and recanalization characteristics of hydrogel microspheres with polyzene-F as polymer coating. Cardiovascular Stampfl S, Stampfl U, Bellemann N, Sommer CM, Thierjung H, Radeleff B, Lopez-Benitez R, Berger I, Kauffmann GW, Richter GM: and interventional radiology 2008, 31:799-806. 9
  - embolization using narrow-size calibrated embozene microspheres. Cardiovascular and interventional radiology 2011, 34:295-305. Stampfl U, Radeleff B, Sommer C, Stampfl S, Dahlke A, Bellemann N, Kauczor H-U, Richter GM: **Midterm results of uterine artery** 20.
- leiomyomas with polyzene F-coated hydrogel microspheres: Initial experience. Journal of Vascular and Interventional Radiology Smeets AJ, Nijenhuis RJ, van Rooij WJ, Lampmann LE, Boekkooi PF, Vervest HA, De Vries J, Lohle PN: Embolization of uterine 21.
- Kalmar PI, Leithner A, Ehall R, Portugaller RH: Is embolization an effective treatment for recurrent hemorrhage after hip or knee arthroplasty? Clinical Orthopaedics and Related Research® 2016, 474:267-271. 22.
- embolization as a treatment for mild to moderate radiographic knee osteoarthritis resistant to conservative treatment. Journal of Okuno Y, Korchi AM, Shinjo T, Kato S, Kaneko T: Midterm clinical outcomes and MR imaging changes after transcatheter arterial Vascular and Interventional Radiology 2017, 28:995-1002.
- Ayis S, Dieppe P: **The natural history of disability and its determinants in adults with lower limb musculoskeletal pain.** The Journal of rheumatology 2009, 36:583-591. 24.
  - Dominick KL, Ahern FM, Gold CH, Heller DA: Health-related quality of life and health service use among older adults with osteoarthritis. Arthritis Care & Research 2004, 51:326-331. 25.

- lkeda K, Nakagomi D, Sanayama Y, Yamagata M, Okubo A, Iwamoto T, Kawashima H, Takahashi K, Nakajima H: **Correlation of** radiographic progression with the cumulative activity of synovitis estimated by power Doppler ultrasound in rheumatoid arthritis: difference between patients treated with methotrexate and those treated with biological agents. The Journal of
- Pap T, Distler O: Linking angiogenesis to bone destruction in arthritis. Arthritis & Rheumatism 2005, 52:1346-1348.

rheumatology 2013, 40:1967-1976.

- Rabin R, Charro Fd: EQ-SD: a measure of health status from the EuroQol Group. Annals of medicine 2001, 33:337-343.
- Riddle DL, Jiranek WA, Hull JR: Validity and reliability of radiographic knee osteoarthritis measures by arthroplasty surgeons. Orthopedics 2013, 36:e25-e32. 27. 28. 29.
- a new adverse event classification by the society of interventional radiology standards of practice committee. Journal of Vascular Khalilzadeh O, Baerlocher MO, Shyn PB, Connolly BL, Devane AM, Morris CS, Cohen AM, Midia M, Thornton RH, Gross K: Proposal of and Interventional Radiology 2017, 28:1432-1437. e1433. 30.
  - Casella, G. (1986). Refining binomial confidence intervals. The Canadian Journal of Statistics, 14, 113--129 31.
- Padia SA et al. Genicular Artery Embolization for the Treatment of Symptomatic Knee Osteoarthritis. JB JS Open Access. 2021 Oct-Dec; 6(4): e21.00085.)

### 19 Attachments

These documents are relevant to the protocol, but they are not considered part of the protocol. They are stored and modified separately. As such, modifications to these documents do not require protocol amendments.

Attachment 1\_Embozene Derections for use (DFU)
Attachment 2\_Embozene FDA K180102
Attachment 3\_Embozene FDA\_K141209
Attachment 4\_RedCap eCRF
Attachment 5\_Study Brochure
Attachment 6\_Recruitment sample subject direct email notification
Attachment 7\_Telephone Recruitment Script
Attachment 8\_FDA-3500A
Attachment 9\_IRB OA Consent\_V0.1\_07.08.2019